

# **Table of Contents**

| 1.0 INTRODUCTION | 3 |
|----------------------------------------------------------------|----|
| 2.0 BRIEF OVERVIEW OF THE STUDY PROTOCOL | 3 |
| 3.0 STUDY STAFF RESPONSIBILITIES | 3 |
| 4.0 STUDY FLOW DIAGRAM | |
| Figure 1: Study Flow Diagram | |
| 5.0 RECRUITMENT AND RETENTION | |
| 5.1 Screening and Eligibility Criteria | |
| 5.2 Screening Log | |
| 5.3 ELIGIBILITY CRITERIA | |
| 6.0 INFORMED CONSENT | |
| 7.0 STUDY INTERVENTION | 5 |
| 8.0 RANDOMIZATION | 5 |
| 9.0 BLINDING AND UNBLINDING (MASKING AND UNMASKING) | 8 |
| 10.0 SAFETY REPORTING | |
| 11.0 STUDY COMPLIANCE | |
| 12.0 DATA COLLECTION AND STUDY FORMS | |
| 12.1 Participant Data | |
| 12.2 Study Forms | |
| 12.3 General Instructions for Completing Forms | |
| 12.4 Data Flow | |
| 12.5 Administrative Forms | 9 |
| 12.6 Retention of Study Documentation | 9 |
| 13.0 DATA MANAGEMENT | |
| 13.1 External Data | |
| 13.2 Quality Control Procedures | 9 |
| 14.0 CONCOMITANT MEDICATIONS | |
| 15.0 DATA AND SAFETY MONITORING ACTIVITIES | |
| 15.1.1 Participant Notification | 10 |
| 15.1.2 Confidentiality Procedures | 10 |
| 16.0 MOP MAINTENANCE | |
| APPENDIX A: IRB-APPROVED STUDY PROTOCOL | 12 |
| APPENDIX B: INFORMED CONSENT DOCUMENTS AND HIPAA AUTHORIZATION | 50 |
| APPENDIX C: MOD MODIFICATIONS LOC | 60 |

#### **1.0 Introduction**

We will measure COVID-19 related preventative health behaviors, including COVID-19 vaccinations, in the Contra Costa County, CA Medicaid managed care population. Our goal is to test ways to increase COVID-19 vaccination uptake. Our hypothesis is that as a result of financial, cultural, or access issues, among other things, vaccinations and other preventative health behaviors are too low from a public health standpoint, meaning relative to virus exposure and the potential adverse consequences of infection in low-income and racial/ethnic minority populations. Furthermore, we hypothesize that small financial incentives and other low-cost behavioral nudges can be used to reduce disparities, increasing vaccination rates and other behaviors known to mitigate the spread of the virus.

#### 2.0 Brief Overview of the Study Protocol

Approximately 10,000 adult subjects will be recruited from the Contra Costa Health Plan (CCHP) via baseline survey. Subjects who complete the baseline survey will be randomized to the following arms:

- 1. Control Arm (n=2,500)
- 2. Informational Arm: no information/emotional message vs. safety and effectiveness information vs. information on consequences of going unvaccinated, race and/or gender concordant or discordant [7,500]

Each of these arms will be interacted with a financial incentive of \$10 (N=2,500) or \$50 (N=2,500) and, separately with a convenient link to the county public vaccine appointment scheduling system highlighted for participants (N=5,000).

The above treatments are designed to test the role of the following on vaccine take-up:

- Financial incentives [N=5,000] vs. no financial incentives [N=5,000]
  - o 2,500 will be randomized to a \$10 incentive and 2,500 to a \$50 incentive
- Convenient scheduling link highlighted [N=5,000] vs. not [N=5,000]
- Messaging [N=7,500] vs not [2,500]
  - Message type: emotion [N=2,500] vs. safety and effectiveness [N=2,500]
     vs. consequences of not vaccinating [N=2,500]
- Race concordant [N=2,500] vs. race discordant messenger [N=2,500]
- Gender concordant [N=2,500] vs. gender discordant messenger [N=2,500]

We will obtain survey data on preventative health behaviors, including mask-wearing, hand washing, and willingness to vaccinate. We will obtain EMR data on vaccine take-up.

#### 3.0 Study Staff Responsibilities

Pilot PI Jacobson will have ultimate responsibility for the study's design and implementation. She will be supported by Other Significant Contributors Tom Chang and Manisha Shah. Jacobson will develop all study materials, including this MOP. She will be

responsible for monitoring and reporting adverse events (AEs), serious adverse events (SAEs), and other issues per the terms of the relevant Data and Safety Monitoring Plan (DSMP). She will obtain informed consent and HIPAA authorization from all subjects; recruit and randomize subjects; receive EMR data from CCHS; following the procedures in this MOP and the IRB-approved protocol; and report any protocol deviations to the IRB and other relevant parties. She will be responsible for protecting subjects' rights on a daily basis. She will oversee all data management procedures and quality control procedures.

Collaborator Rajiv Pramanik of Conta Costa Health System (CCHS) will facilitate subject contacts and sharing of EMR data. CCHS will provide data on eligible CCHP members and will be responsible for screening members for eligibility.

## 4.0 Study Flow Diagram

Figure 1: Study Flow Diagram



#### 5.0 Recruitment and Retention

A random sample of eligible CCHP members will be invited to participate in the study via email, mail, and/or text. We aim to recruit 10,000 subjects and recruitment will continue until we have reached 10,000 baseline survey responses.

We will provide gift cards for baseline survey completion (\$5 or \$25, depending on survey take-up). In addition, respondents will be entered into a raffle for \$250 gift cards.

#### 5.1 Screening and Eligibility Criteria

CCHS will provide a list of eligible members and will be responsible for eligibility screening. Pilot PI Jacobson will not be responsible for eligibility screening. See 5.3 for Eligibility Criteria.

### 5.2 Screening Log

As screening will not be performed by Pilot PI Jacobson or her academic study team, this group will not maintain a screening log. Collaborator Pramanik will maintain documentation of eligibility determinations.

#### 5.3 Eligibility Criteria

Eligible subjects are adult CCHP members with no previous COVID-19 vaccination history and no contraindications to COVID-19 vaccination, as determined in CCHP medical staff.

#### **6.0 Informed Consent**

Informed consent will be obtained during the baseline survey to recruit subjects. The IRB-approved consent documents are attached as an appendix.

#### 6.1 HIPAA Authorization

Personal health information (PHI) will be obtained in keeping with the Health Insurance Portability and Accountability Act (HIPAA). The IRB approved a partial HIPAA waiver for purposes of study participant recruitment. The study outcome, COVID-19 vaccination, is PHI. The IRB-approved HIPAA authorization form is attached as an appendix.

#### 7.0 Study Intervention

Subjects in treatment arms will receive interventions:

- Financial incentives [N=5,000] vs. no financial incentives [N=5,000]
  - 2,500 will be randomized to a \$10 incentive and 2,500 to a \$50 incentive
- Convenient scheduling link highlighted [N=5,000] vs. not [N=5,000]
- Messaging [N=7,500] vs not [2,500]
  - Message type: emotion [N=2,500] vs. safety and effectiveness [N=2,500] vs. consequences of not vaccinating [N=2,500]
- Race concordant [N=2,500] vs. race discordant messenger [N=2,500]
- Gender concordant [N=2,500] vs. gender discordant messenger [N=2,500]

#### 8.0 Randomization

We will stratify our sample based on based on race/ethnicity and age-group. Randomization will be performed in the RedCAP system. In practice, the randomization will divide the sample into 60 possible conditions:

- 1. Control [N=625]
- 2. Control x \$10 financial [N=312.5]
- 3. Control x \$50 financial [N=312.5]

- 4. Control x link [N=625]
- 5. Control x \$10 financial x link [N=312.5]
- 6. Control x \$50 financial x link [N=312.5]
- 7. No information/Emotional (language concordant) [N=625]
- 8. No information/Emotional (language concordant) x \$10 financial [N=312.5]
- 9. No information/Emotional (language concordant) x \$50 financial [N=312.5]
- 10. No information/Emotional (language concordant) x link [N=625]
- 11. No information/Emotional (language concordant) x \$10 financial x link [N=312.5]
- 12. No information/Emotional (language concordant) x \$50 financial x link [N=312.5]
- 13. Safety and effectiveness (race concordant, male) [N=156.25]
- 14. Safety and effectiveness (race concordant, male) x \$10 financial incentive [N=78.125]
- 15. Safety and effectiveness (race concordant, male) x \$50 financial incentive [N=78.125]
- 16. Safety and effectiveness (race concordant, male) x link [N=156.25]
- 17. Safety and effectiveness (race concordant, male) x \$10 financial incentive [N=78.125]
- 18. Safety and effectiveness (race concordant, male) x \$50 financial incentive [N=78.125]
- 19. Safety and effectiveness (race concordant, female) [N=156.25]
- 20. Safety and effectiveness (race concordant, female) x \$10 financial incentive [N=78.125]
- 21. Safety and effectiveness (race concordant, female) x \$50 financial incentive [N=78.125]
- 22. Safety and effectiveness (race concordant, female) x link [N=156.25]
- 23. Safety and effectiveness (race concordant, female) x \$10 financial incentive x link [N=78.125]
- 24. Safety and effectiveness (race concordant, female) x \$50 financial incentive x link [N=78.125]
- 25. Safety and effectiveness (race discordant, male) [N=156.25]
- 26. Safety and effectiveness (race discordant, male) x \$10 financial incentive [N=78.125]
- 27. Safety and effectiveness (race discordant, male) x \$50 financial incentive [N=78.125]
- 28. Safety and effectiveness (race discordant, male) x link [N=156.25]
- 29. Safety and effectiveness (race discordant, male) x financial incentive x link [N=78.125]
- 30. Safety and effectiveness (race discordant, male) x financial incentive x link [N=78.125]
- 31. Safety and effectiveness (race discordant, female) [N=156.25]
- 32. Safety and effectiveness (race discordant, female) x \$10 financial incentive [N=78.125]

- 33. Safety and effectiveness (race discordant, female) x \$50 financial incentive [N=78.125]
- 34. Safety and effectiveness (race discordant, female) x link [N=156.25]
- 35. Safety and effectiveness (race discordant, female) x \$10 financial incentive x link [N=78.125]
- 36. Safety and effectiveness (race discordant, female) x \$50 financial incentive x link [N=78.125]
- 37. Consequences of going unvaccinated (race concordant, male) [N=156.25]
- 38. Consequences of going unvaccinated (race concordant, male) x \$10 financial incentive [N=78.125]
- 39. Consequences of going unvaccinated (race concordant, male) x \$50 financial incentive [N=78.125]
- 40. Consequences of going unvaccinated (race concordant, male) x link [N=156.25]
- 41. Consequences of going unvaccinated (race concordant, male) x \$10 financial incentive x link [N=78.125]
- 42. Consequences of going unvaccinated (race concordant, male) x \$50 financial incentive x link [N=78.125]
- 43. Consequences of going unvaccinated (race concordant, female) [N=156.25]
- 44. Consequences of going unvaccinated (race concordant, female) x \$10 financial incentive [N=78.125]
- 45. Consequences of going unvaccinated (race concordant, female) x \$50 financial incentive [N=78.125]
- 46. Consequences of going unvaccinated (race concordant, female) x link [N=156.25]
- 47. Consequences of going unvaccinated (race concordant, female) x \$10 financial incentive x link [N=78.125]
- 48. Consequences of going unvaccinated (race concordant, female) x \$50 financial incentive x link [N=78.125]
- 49. Consequences of going unvaccinated (race discordant, male) [N=156.25]
- 50. Consequences of going unvaccinated (race discordant, male) x \$10 financial incentive [N=78.125]
- 51. Consequences of going unvaccinated (race discordant, male) x \$50 financial incentive [N=78.125]
- 52. Consequences of going unvaccinated (race discordant, male) x link [N=156.25]
- 53. Consequences of going unvaccinated (race discordant, male) x \$10 financial incentive x link [N=78.125]
- 54. Consequences of going unvaccinated (race discordant, male) x \$50 financial incentive x link [N=78.125]
- 55. Consequences of going unvaccinated (race discordant, female) [N=156.25]
- 56. Consequences of going unvaccinated (race discordant, female) x \$10 financial incentive [N=78.125]
- 57. Consequences of going unvaccinated (race discordant, female) x \$50 financial incentive [N=78.125]

- 58. Consequences of going unvaccinated (race discordant, male) x link [N=156.25]
- 59. Consequences of going unvaccinated (race discordant, male) x \$10 financial incentive x link [N=78.125]
- 60. Consequences of going unvaccinated (race discordant, male) x \$50 financial incentive x link [N=78.125]

Randomization assignments will be documented for future reference.

#### 9.0 Blinding and Unblinding (Masking and Unmasking)

There is no scope for masking in this study. Subjects will know that treatment they have received, if any. We will not mask care providers or outcomes assessors.

#### 10.0 Safety Reporting

Per our DSMP, we will be unable to observe AEs and SAEs in our survey and EMR data.

Routine monitoring of EMR data for AEs and SAEs will not be conducted.

However, if the research team becomes aware through other channels of a specific event, the report will immediately be relayed to the PIs.

The PI will determine whether the event constitutes an AE or SAE, and classify any AEs or SAEs on their severity, expectedness, and relatedness, as above. The PI will consult with a qualified clinician as necessary to make such determinations. Affected subjects will be advised to visit a local, qualified medical practitioner.

Unexpected SAEs will be reported to the Safety Officer (SO), IRB, and NIA within 48 hours of the study's knowledge, and summarized in periodic electronic reports to the SO.

Any unanticipated problem, defined as an issue related to the research that suggests the research places participants or others at greater risk than was expected, will be reported to NIA and the SO within 48 hours of the study's knowledge. Reporting will occur within 24 hours if the problem involves death. The report will include a plan to correct the problem and prevent its reoccurrence.

Any SAEs related to the study and any unanticipated problems will also be promptly reported to the sIRB.

#### 11.0 Study Compliance

Protocol deviations for this study, while exceedingly unlikely, could include randomizing an ineligible participant; obtaining incomplete or inadequate informed consent; administering the wrong treatment to a subject; or failing to keep the IRB protocol up to date.

Any deviations that impact participant safety will be reported to NIA and the SO within 24 hours of occurrence, or as soon as they are discovered. All other deviations will be

captured in routine reports to NIA and the SO. All deviations will be reported to the sIRB of Record in accordance with local policies and captured in the protocol deviations log in the appendix of this MOP.

## 12.0 Data Collection and Study Forms

## 12.1 Participant Data

Individual-level survey data, EMR data, and randomization information will be maintained electronically by the study team. Survey data will be received directly by the study team. EMR data will be transmitted from CCHS to the study team.

## 12.2 Study Forms

There are no study-specific forms for this study.

#### 12.3 General Instructions for Completing Forms

Not applicable.

#### 12.4 Data Flow

Data, which will include PHI, will be stored on secure servers only available to the research team. Coded data will be used for analysis and will be stored separately from the identifiable data.

#### 12.5 Administrative Forms

We will use the Adverse Event Form and Serious Adverse Event Form from the NIA Clinical Research Study Investigator's Toolbox to record any AEs or SAEs.

#### 12.6 Retention of Study Documentation

Participant data will be retained by the study team for at least the NIH minimum of three years. We have no plans for data destruction at this time. Informed consent will be included in the baseline survey data and maintained indefinitely.

#### 13.0 Data Management

#### 13.1 External Data

The study team will receive data from CCHS on eligible CCHP members and on enrolled subjects' vaccine outcomes. These data transfers will rely on Box.com, which encrypts the data during transfer and at rest. USC and CCHS will execute appropriate data use agreement(s) before transferring any data.

#### 13.2 Quality Control Procedures

The study team will review data from CCHS, as well as survey data, as soon as possible after receipt. The team will perform standard data quality checks, to include flagging missing, out-of-range, or illogical data.

#### **14.0 Concomitant Medications**

Not applicable.

#### 15.0 Data and Safety Monitoring Activities

#### 15.1 Study Completion and Close-Out Procedures

At close-out, Pilot PI Jacobson will ensure that all required data has been received and that all data and analysis files are organized and accessible for review. She will ensure that all required study information has been reported to the NIA and other funders. She will notify the IRB of Record of the study's completion and retain a copy of this notification. Finally, she will prepare a report summarizing the study's conduct.

#### 15.1.1 Participant Notification

We do not plan to notify subjects or their health providers of the results of the study.

## 15.1.2 Confidentiality Procedures

Data will be stored securely as described in 12.4 and 13.1 above. Data will be accessed only by staff with a legitimate need. All staff will be properly trained in human subjects research practices and appropriately supervised.

If computers are used to store and/or analyze clinical data, the investigator should address elements of computer security to ensure that the data remain confidential. These elements include but are not limited to: utilization of computer and system passwords, user security training, system testing and verification, and routine system backups to prevent any loss of electronic data.

## 16.0 MOP Maintenance

Each page of the MOP is numbered, dated, and includes a version number. Modifications are logged in the appendix.



## APPENDIX A: IRB-Approved Study Protocol and 06/01/2021 Amendment

UP-21-00030 - COVID-19 and Preventive Health Behaviors

4/29/21, 8:48 AM

Version: 1.4

Application Version Date: 4/28/2021

| 1. Project Identification and Abstr | ac | :t |
|-------------------------------------|----|----|
|-------------------------------------|----|----|

| 1. 1 | roject identification and Abstract |
|---|---|
| 1.1. | Type of Submission: |
| | Research Protocol or Study on Human Subjects |
| | Grant/Contract Only |
| | Use of Humanitarian Use Device (Not Research) |
| | Rely on another IRB (Ceded) |
| 1.2. | Full Title of Research Protocol<br>COVID-19 and Preventive Health Behaviors in at-Risk Medicaid Populations |
| 1.3. | Short Title<br>COVID-19 and Preventive Health Behaviors |
| 1.4. | Abstract: Provide a simple explanation of the study and briefly address (in 1 to 2 sentences) each of the following points: rationale; intervention; objectives or purpose; study population or sample characteristics; study methodology; description of study arms (if appropriate); study endpoints or outcomes; follow-up; statistics and plans for analysis. In this work, we are partnering with Contra Costa Health Services (CCHS), the department of health in Contra Costa County, CA, to measure COVID-19 related preventive health behaviors, including COVID-19 vaccinations, in the county Se Medicaid managed care population and test ways to increase COVID-19 vaccine uptake. Our hypothesis is that, as a result of financial, cultural or access issues, among other things, vaccinations and other preventive health behaviors are too low from a public nealth standpoint, meaning relative to virus exposure and the potential adverse consequences of infection in low-income and racial/ethnic minority populations. Furthermore, we hypothesize that small financial incentives and other low-cost behavioral mudges can be used to reduce disparities, increasing vaccination rates and other behaviors known to mitigate the spread of the virus. |

1.5. \* Select which IRB you are requesting review from:

| O USC - Biomedical IRB |
|------------------------------------------|
| USC - Social Behavioral IRB |
| CHLA - Institutional Review Board (CHLA) |

Select "USC & Biomedical" if you are conducting biomedical research activities which fall under FDA jurisdiction (drugs, devices, etc.).

Select "USC & Social Behavioral" if you are conducting social behavioral research activities (community/field-based research such as survey and interview procedures, etc. that are not FDA regulated.).

NOTE: IRBAs and designated reviewers (Chairs, Vice Chairs, etc.) are currently assigned to review applications based on the type of research conducted. Selecting the incorrect board may result in a delay of the review process; and the application may be returned for the correct review board to be selected.

1.6. \*To the investigator's knowledge, does the Institution have financial and/or intellectual property interests in the sponsor or the products used in this project?

An institutional conflict may occur when a financial interest of the institution has the potential to bias the outcome of research conducted by its employees or students or to create an unacceptable risk to human subjects.

https://istar.usc.edu/istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.html




#### 2. Study Personnel

#### 2.1. Study Personnel and their roles:

| | Last<br>Name | First<br>Name | Organization | Study<br>Role | Certifications | Obtain<br>Consent | Interact<br>with<br>Participants | Access<br>Identifiable<br>Data | Access<br>to | COVID<br>Attestation<br>(USC<br>Only) |
|---|---|---|---|---|---|---|---|---|---|---|
| View | Jacobson | Mirailla | DAVIS SCHOOL<br>OF<br>GERONTOLOGY | Principal<br>Investigator | HS GCP<br>HIPAA | no | no | yes | | • |
| View | Chang | Tom | MARSHALL<br>SCHOOL OF<br>BUSINESS | Co-<br>Investigator | HS GCP<br>HIPAA | no | no | yes | | • |

#### Who may be included as "key personnel" on an IRB submission?

Key Personnel are individuals who contribute to the scientific development or execution of a project in a substantive, measurable way, whether or not they receive salaries or compensation under the protocol. Individuals who should be named on an IRB application are those who engage in the following:

- a. conducting research through an interaction or intervention with human subjects for research purposes
- b. participating in the consent process by leading it or contributing to it
- directly recording or processing identifiable private information, including protected health information, related to those subjects for the purpose of conducting the research study

#### Who should NOT be listed as key personnel on an IRB submission:

Individuals paid by the institution to perform a service not part of or paid by the research project performing services that are typically performed for non-research purposes or fee for service:

- honest broker
- pharmacy employees dispensing investigations drugs
- hospital employees obtaining blood through a blood draw or collect urine and provide such specimens to investigators as a service
- radiology clinic employees performing chest x-rays and sending results to investigators as a service
- routine laboratory analyses of blood samples for investigators as a commercial service
- · transcription of research study interviews as a commercial service
- not administering any study intervention being tested or evaluated under the protocol

| 2.2. | Is the Principal Investigator a staff member, student, resident, fellow, postdoctoral scholar, other trainee, or visiting |
|---|---|
| | scholar/faculty member at USC/CHLA? |
| | Yes No |

| .5. | Specify the group/organization who has reviewed this study for scientific merit: |
|---|---|
| | Federal Agency (e.g. FDA, NIH, CDC, DOE, NSF, DOJ, etc.) |
| | USC Norris Clinical Investigations Committee |
| | O Doctoral Dissertation Committee |

https://istar.usc.edu/istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.html


| JP-21-00 | 030 - 0 | OVID-19 and Preventive Health Behaviors Other None | 4/29/21, | 8:48 AM |
|---|---|---|---|---|
| 4. | | Specify the other group/organization who has J-PAL North America ding Information | as reviewed this study for scientific merit: | |
| 4.1. | * Wh | at existing or pending support will be used fo | r this study? (check all that apply) | |
| | | Cooperative Group (SWOG, COG, RTOG, etc.) | | |
| | | CTSI | | |
| | | Department of Defense (DOD) Funds | | |
| | | Departmental/Institutional Funds | | |
| | <b>~</b> | Federal Grant/Contract | | |
| | <b>~</b> | Foundation Grant/Contract | | |
| | | Industry | | |
| | | Intramural/Internal Grant | | |
| | | Residual Funds | | |
| | | State or Local Grant/Contract | | |
| | | Subcontract from another institution | | |
| | | No Funding | | |
| | ~ | Other | | |
| | ì | Change of existing/addition of new funding so | urces and agencies will require an amendment. | |
| | | Will you be submitting an Urgent Review red Yes No Will any funds come from the National Instit Yes No | | - |
| 4.2. | proje | | ew by the IRB (i.e., cooperative group grants, umbrella grants, mult<br>it it from the list using the 'Add' button. If the funding source is not<br>ion 4.4. | |
| | Gran | t# Principal Investigator | Grant Title | |
| ttps://ist | ar.usc.e | du/istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/f | romString.html Pag | e 3 of 29 |

There are no items to display

4.2.1. If the grants selected in question 4.2 fund multiple studies, please attach the specific pages of the grant that are relevant to THIS study.

Name Version Modified

There are no items to display

4.4. Add the details of each source of funding for this study.

| Sponsor | Principal Investigator | Type of Funding |
|---|---|---|
| View National Institutes on Aging | Joe Doyle and David Laibson | Federal: Program Project/Multiple Project Grant * |

4.5. For those studies with a related award in the USC award system, Kuali Coeus, please use the "Find Now" button below to relate this study with the award(s):

Related Awards (uncheck checkbox to remove):

| PI PI Last<br>First Name<br>Name | Institutional<br>Proposal<br>Number | USC<br>Award<br>Number | Project Title | Prime<br>Sponsor<br>Name | Sponsor Name | Project<br>Start<br>Date | Co<br>Investigators |
|---|---|---|---|---|---|---|---|
| Mireille Jacobso | n 00220372 | | COVID-19 and Preventive<br>Health Behaviors in at-Risk<br>Medicaid Populations | | Abdul Latif<br>Jameel Poverty<br>Action Lab | 2/1/2021 | |

#### 5. Type of Study Review

5.1. Select the type of review that you are requesting for this study:

| 0 | Full Committee Review |
|---|-----------------------|
| • | Expedited Review |
| 0 | Exempt Review |
| 0 | Coded Specimens/Data |

5.2. Attach the protocol here. All studies require a fully developed protocol. If you have questions contact the IRB office to discuss.

| name | versio | on Woaltlea |
|-------------------------------------|--------|-------------------|
| Amended Protocol - April 2021(0.05) | 0.05 | 4/23/2021 3:26 PM |

A grant proposal is not applicable, and should not be uploaded in lieu of a protocol (template is attached and will also be available on the OPRS website).

Protocol Template: Social-Behavioral

https://istar.usc.edu/istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.html


| JP-21-00030 - | COVID-19 and | Preventive | Health | Behaviors |
|---------------|--------------|------------|--------|-----------|

4/29/21, 8:48 AM

5.3. Attach the sponsor's template informed consent here.

Name Version
There are no items to display

5.4. If any study documents are password protected, enter the passwords here.

Modified

5.5. If there is a sponsor protocol number associated with this file, specify it here:

#### 6. Study Locations

| 6.1. | Identify | the locations | where the | research | activities | described | in this | application | will be | performed | (check al | I that app | ply) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

| USC HSC - | Health | Sciences | Associated | Locations |
|-----------|--------|----------|------------|-----------|
|-----------|--------|----------|------------|-----------|

| ~ | USC UPO | C - University | Park | Associated | Locations |
|---|---------|----------------|------|------------|-----------|
|---|---------|----------------|------|------------|-----------|

| OLII. |
|-------|
| CHL/ |

Other

6.2. Will USC/CHLA serve as the reviewing IRB for the other sites (single IRB model)?

| Yes | ALC: U | No |
|---------|--------|-----|
| <br>165 | | INO |

## 6b. UPC Location(s)

This screen is required if you indicated UPC - University Park Associated Locations (Question 6.1.)

6b.1. UPC Locations (check all that apply and provide detail where indicated):

Location

✓ Campus location (includes ISI and ICT)

Off-campus location

If campus location, please specify:

Davis School of Gerontology

6b.2. If off-campus location, please specify:

#### 6d. Other Sites/Institutions

This screen is required if you indicated that USC/CHLA is the lead institution or is conducting the study at other sites (Question 6.2.1.1. or 6.2.2.).

6d.1. List ALL participating sites below:

| Site Name | Address | Engagement |
|---|---|---|
| View Contra Costa Health Services | 333 C Street, Martinez, CA 94553 | |

https://istar.usc.edu/istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.html


View MIT/JPAL 400 Main Street E19-201 Cambridge, MA 02142 USA

View National Bureau of Economic Research (NBER) 1050 Massachusetts Ave, Cambridge, MA 02138 Engaged

# 9. Methods and Procedures - Selected Descriptors/Community Engaged Research

Note: The list of items below IS NOT an all-inclusive list of methods and procedures available to investigators. The list only includes items that will trigger additional questions specific to areas of research or are necessary for the review process.

| 9.1. | | Study will include: (check all that apply) Data/specimens that will be collected for research purposes | |
|---|---|---|---|
| | ~ | Data/specimens that have been or will be collected for non-rese | earch purposes (e.g., clinical care, student records) |
| | 9.1.1 | . Will anyone in the study team (listed under Section 2.1) had yes No | ave direct in-person interaction with participants? |
| 9.2. | Stud | y Procedures: (check all that apply) | |
| | | Audio/Video Recordings or Photographs | |
| | | Behavioral Observations and/or Behavioral Experimentation | |
| | ~ | Behavioral Interventions | |
| | | Deception | |
| | | Interview/Focus Groups | |
| | | Population-based Field Study | |
| | | Psychophysiological Testing | |
| | ~ | Surveys/Questionnaires/Psychometric Testing | |
| | | Approved/Investigational Devices | |
| | | Biohazardous Substances (e.g. fresh tissue or tissue fluids, info<br>of biological material) | ectious agents, microorganisms, recombinant DNA, or shipment |
| | | Blood Collection | |
| | | Creation of a Data or Tissue Repository | |
| | | Magnetic Resonance Imaging (MRI) | |
| | | Stem Cells or Cell-Based Therapy | |

9.3. Is this a clinical trial? [The NIH defines a clinical trial as a prospective research study to evaluate the effects of one or more interventions on health-related biomedical or behavioral outcomes.]

https://istar.usc.edu/istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.html


| JP-21-00030 - | COVID-19 and | Preventive | Health Be | ehaviors |
|---------------|--------------|------------|-----------|----------|

4/29/21, 8:48 AM

| Yes | No No |
|-----|-------|
| 103 | ) INU |

Clinical Trials must be registered on clinicaltrials.gov. All study personnel on studies meeting the NIH definition of clinical trials are required to satisfy the Good Clinical Practice (GCP) education requirement.

9.5. Will data from this study be subject to the NIH Genomic Data Sharing (GDS) policy?

Yes No

9.6. Does your study involve community-engaged research (community-engaged research addresses community needs and involves the community in research plan, conduct of study, etc)?

Yes No

9.6.1 How is the community involved? (select all that apply)

Community Advisory Board established for this study provides input Study results are/will be disseminated to the community

9.7. Will data from this research be submitted to the US Food and Drug Administration or will data be held for inspection by the FDA?

Yes No

#### 10. Characteristics of the Study Subject Population

- 10.1. What is the maximum number of subjects you plan to recruit for this site? (Integer values only)
  - 10.1.1. If this is a multi-site study, indicate the projected total subject accrual. (Integer values only)
  - 10.1.2. If necessary, provide further explanation of accrual goals for all subject populations. Baseline survey enrollment is targeted at 10,000.
  - 10.3.1. If there are any age, ethnic, language, or gender-based exclusion criteria, please provide justification. Ages 18 and over because they make health care decisions for themselves.

To analyze the issue of race concordance on vaccine take-up, we will focus on White, Black, and Latinos of any race. We will need to exclude racial minorities that are too small a share of the CCHP population to allow us to make inferences about race concordance. As a result, we exclude CCHP members identified as American Indian/Alaska Native and Hawaiian/Pacific Islanders as each group accounts for less than 1% of enrollees. We will also exclude Asians, a group that is very heterogenous generally and in Contra Costa specifically. When grouped together as a single �race, � Asians account for about 15% of the CCHP population. However, that group is comprised of populations that are both linguistically and culturally quite distinct. In particular, about a third of the �Asian � group is Filipino, a third Vietnamese, 25% Mandarin-speaking Chinese, 20% Cantonese-speaking Chinese, 15% Punjabi-speaking Indian, 10% Laotian, 10% Korean, and so on. As such, we do not think these populations can credibly be treated as one group for the purposes of studying race concordance and yet each group is individually too small to consider alone.

https://istar.usc.edu/istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.html


| 13. | Methods | and | Procedures | ; | Collection | of | Data/ | Spe | ecim | ens |
|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|

| 13.1. | Does the study involve collection of data, records or specimens from deceased individuals? |
|---|---|
| | ○ Yes ● No |

13.2. Attach a copy of the Data Collection forms you intend to use to access and record data for research purposes. Data Collection forms include a summary of the variables to be recorded from the original source.

| Name | Version Modified | |
|----------------------|------------------|---------|
| Secondary data(0.01) | 0.01 1/7/2021 : | 3:19 PM |

13.2.1. Will you be obtaining data from a clinical data warehouse (such as the CDW at Keck or LA County)?

| Yes | 0 | No |
|-----|---|----|

- 13.3. Describe the method of collection for the records/specimens and how the data/specimens will be analyzed.
  - 13.3.a. Specify the number of records/specimens you expect to use: (This is a deprecated field only used for existing studies.) 10000
- 13.4. Describe the method(s) by which subject records will be identified.

# 21. Methods and Procedures - Surveys/Questionnaires/Psychometric Testing

This screen is required if you indicated the use of Surveys, Questionnaires, or Psychometric Testing (Question 9.2.)

21.2. Attach copies of all measures/instruments that will be used for this study.

| Name | Version Modified |
|-----------------------|-----------------------|
| Baseline survey(0.01) | 0.01 1/7/2021 3:24 PM |

#### 22. Special Subject Populations

| 22.1. | Indic | cate any special subject populations you intend or expect to enroll in the research: (che | ck all that apply) |
|---|---|---|---|
| | | Healthy Volunteers | |
| | | Employees or Students | |
| | | Adults not Competent to Consent (or likely to lose the capacity to consent during the study) | |
| | ~ | Non-English Speaking Populations | |
| | | Minors (subjects under 18 years of age) | |
| | | Pregnant Women / Human Fetuses | |

https://istar.usc.edu/istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.html


| 21-00030 | - COVID-19 and Preventive Health Behaviors | 4/29/21, 8:48 |
|---|---|---|
| | Neonates (infants under 30 days old) | |
| | Prisoners/Detainees | _ |
| | Wards | |
| - | Military Personnel | - |
| | None of the above | |
| Wildell Co. | Special Subject Populations - Non-English Speaking | to the second se |
| | Describe how you will communicate with non-English speaking participants for the purp consent, permission, and or assent. (check all that apply) | , |
| | Translated full consent, permission, and/or assent forms (incl. information sheets) by an authorized interpreter | with verbal interpretation |
| | Translated short forms with verbal interpretation by an authorized interpreter | |
| | Other | |
| 22d.2. | If the study will likely include subjects and families for whom Spanish is the primary lan documents must be translated into Spanish. Select the method of translation. Investigator/Sponsor will provide the IRB with a translation of the approved conser | |
| | Request that the IRB office translate (HSIRB Only) | |
| | Please be advised that a Certificate of Translation may be required if an outside translator is u | ised. |
| | f the research will primarily include subjects who speak a language other than English o<br>consent documents should be translated into that language. Indicate the languages and | |
| | Language Translation Method | |
| | There are no items to display | |
| 00 0 | Andr December | |
| OWEND AND AND ADDRESS OF THE PERSON ADDRESS OF THE PERSON AND ADDRESS OF THE PERSON ADDRESS OF | tudy Resources Describe the time the investigators have available to conduct and complete the research | and justify that it is |
| | ufficient. Please check-off the items that apply to this study. | |
| | Employed interns, residents, fellows, or postdocs with dedicated time to conduct this resear | |
| - | _ | arch. |
| | Employed faculty and or staff with dedicated time to conduct this research. | arch. |

| ээ | 80 – COVID-19 and Preventive Health Behaviors | 4/29/21, |
|---|---|---|
| | Volunteers | |
| | Other | |
| | Describe the staff and justify their qualifi | cations. Please check-off the items that apply to this study. |
| | All biomedical investigators are privile | ged and credentialed to perform the study activities in the study locations. |
| | All study staff are trained and crede | entialed to perform the duties assigned to them. |
| | All study staff have fulfilled the training | mandated by their respective departments or institutions. |
| | Other | |
| | | ney are adequate.<br>nave funds to hire a research manager and a research assistant to help implemen |
| | Subject Recruitment and | Informed Consent |
| | | e local site (check a box only if your site will control the use or distribution |
| | - | e local site (check a box only if your site will control the use or distribution |
| | Recruitment Tools that will be used by the of the recruitment tool): (check ALL that a | e local site (check a box only if your site will control the use or distribution |
| | Recruitment Tools that will be used by the of the recruitment tool): (check ALL that a Brochures | e local site (check a box only if your site will control the use or distribution |
| | Recruitment Tools that will be used by the of the recruitment tool): (check ALL that a Brochures Clinical Data Warehouse | e local site (check a box only if your site will control the use or distribution |
| | Recruitment Tools that will be used by the of the recruitment tool): (check ALL that a Brochures Clinical Data Warehouse Email/Electronic Mailing Lists | e local site (check a box only if your site will control the use or distribution |
| | Recruitment Tools that will be used by the of the recruitment tool): (check ALL that a Brochures Clinical Data Warehouse Email/Electronic Mailing Lists Flyers | e local site (check a box only if your site will control the use or distribution pply) - |
| | Recruitment Tools that will be used by the of the recruitment tool): (check ALL that a Brochures Clinical Data Warehouse Email/Electronic Mailing Lists Flyers Letters | e local site (check a box only if your site will control the use or distribution pply) - |
| | Recruitment Tools that will be used by the of the recruitment tool): (check ALL that a Brochures Clinical Data Warehouse Email/Electronic Mailing Lists Flyers Letters Newspaper/Magazine Advertisements | e local site (check a box only if your site will control the use or distribution pply) - |
| | Recruitment Tools that will be used by the of the recruitment tool): (check ALL that a Brochures Clinical Data Warehouse Email/Electronic Mailing Lists Flyers Letters Newspaper/Magazine Advertisements Radio/Television Announcements | e local site (check a box only if your site will control the use or distribution pply) - |
| | Recruitment Tools that will be used by the of the recruitment tool): (check ALL that a Brochures Clinical Data Warehouse Email/Electronic Mailing Lists Flyers Letters Newspaper/Magazine Advertisements Radio/Television Announcements Subject or Participant Pools | e local site (check a box only if your site will control the use or distribution pply) - |
| | Recruitment Tools that will be used by the of the recruitment tool): (check ALL that as a Brochures Clinical Data Warehouse Email/Electronic Mailing Lists Flyers Letters Newspaper/Magazine Advertisements Radio/Television Announcements Subject or Participant Pools Telephone Scripts | e local site (check a box only if your site will control the use or distribution pply) - |


| -000 | 30 - CO\ | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Vone | of the | above | | | | | | | | | | | | | | | | |
| | 24.1.1 | | ease s<br>xt | pecify: | | | | | | | | | | | | | | | | |
| | 24.1.2 | | | | ou will b<br>e a list o | | | | infor | matior | 1: | | | | | | | | | |
| 2. | | | | | uitment<br>sed at th | | | | | | | | o not | attach | any ad | dvertis | sing o | r recru | itment | |
| | Name | | at wiii i | or be u | seu at tr | ie iocai s | | | n Moc | | local | 3110.) | | | | | | | | |
| | | | itment | email te | ext(0.02) | | | 02 | | 8/2021 | 4:38 F | PM | | | | | | | | |
| 3. | Inform | ned ( | onsen | t and W | /aivers: | | | | | | | | | | | | | | | |
| | ** Ple | ase r | ote th: | t child | assent a | and nar | ental ne | rmis | sion v | will he | addn | hasse | l on s | uhser | went | nane | s Do | not co | mnlete | |
| | | | | | estions | | | | | | | | | | • | | | | • | |
| | Checl | the: | type(s) | of con | sent or | waiver ( | of cons | ent p | lanne | d for t | his st | udy: ( | (chec | k ALL | that ap | oply) | | | | |
| | _ | | | | sent or<br>sent (pa | | | | | | | | | | that ap | oply) | | | | |
| | <b>V</b> | <b>Writt</b><br>Altera | en/sigr | ed con | | a <b>rticipa</b> n | nts will s | si <b>gn</b> a | an inf | ormed | cons | ent d | ocun | ent) | | | of the | e basic | require | d |
| | | Writt<br>Altera | en/sigr | ed con<br>the eler<br>consent | sent (pa | articipan<br>consent<br>altered o | nts will s<br>(particip<br>r waived | s <b>ign</b> a<br>pants | an inf | ormed | onsen | ent de | ocun<br>umen | n <b>ent)</b><br>t, but c | ne or | more | | | | d |
| | | Writt<br>Altera<br>elema<br>Waiva | en/sigr<br>tion of<br>ents of | ed con<br>the eler<br>consent<br>ned info | sent (pa<br>ments of<br>will be a | consent<br>altered o | ts will s<br>(particip<br>r waived | sign a | an inf<br>will s | ormedign a c | onsen | ent docu | ocun<br>umen | n <b>ent)</b><br>t, but c | ne or | more | | | | d |
| 7. | Attacinfor | Writt Altera Altera Waive Waive | en/sigr<br>tion of<br>ents of<br>er of sig<br>er of co<br>pies of | the eler<br>consent<br>ned info<br>nsent (p | sent (pa<br>ments of<br>will be a<br>ormed co | consent (ints will not consent to consent to consent to consent to consent to adden | (participate of the decument of the as document of the as document of the the decument of the the decument of the the decument of the | sign and some si | an inf will s sent d o sign (s), in cable | ign a cocume | onsen | t docu | ocumenthe signsent | nent) t, but constured document | e section<br>ent)<br>tatem<br>dy. Th | more | ill be p | provide<br>w | ed) | |
| 7. | Attacinfor | Writt Altera Altera Waive Waive Ch cccmati | en/sign<br>ents of<br>er of sign<br>er of co<br>pies of<br>on/find<br>at or pa | the eler<br>consent<br>med info<br>nsent (p | sent (pa<br>ments of<br>will be a<br>participar<br>formed of<br>consen<br>permiss | consent (ints will not consent to consent to consent to consent to consent to adden | (participate of the decument of the as document of the as document of the the decument of the the decument of the the decument of the | sign and some si | an inf will s sent d o sign (s), in cable | ign a cocume | onsenonsent with given tion solil bed. | t docu | ocumen he signature sent | nent) t, but of nature docum any s is stu | e section<br>ent)<br>tatem<br>dy. Th | more ons w ents | ill be p | provide<br>w | ed) | |
| 7. | Attacinfor | Writt Altera Waive Waive Ch ccrmati asse e Con | en/sigr<br>tion of<br>ents of<br>er of sig<br>er of co<br>pies of<br>on/find<br>at or pa | the elerconsent ined information (processed for the information of the | sent (pa<br>ments of<br>will be a<br>participar<br>formed of<br>consen<br>permiss | consent (ints will not consent to addentify addentify addentify addentify and a consent to addentify addentification addentify addentify addentify addentify addentify addentify addentify addentification add | r (partici)<br>r (partici)<br>r waived<br>nformed<br>ot be as<br>docum<br>da (as a<br>uments | pants cons ked t ents applic that | an infi<br>will s<br>seent d<br>o sign<br>(s), in<br>cable) | ign a cocume | onsennt with given stion servill be | t docu<br>t docu<br>nout th<br>a cons<br>heets<br>used | ocum umen ne sig sent i, and l in th | nent) t, but constructed any sany suis stu | e section<br>ent)<br>tatem<br>dy. Th | more ons w ents ents se | ill be p | provide<br>w | ed) | |
| 7. | Attacinfor any Nam | Writt Altera Altera Waive Waive Con HIP, | en/sigr<br>tition of<br>ents of ents | the elerconsent in the information of the informati | sent (pa | consent (ints will not consent to addentify addentification addentification addentify addentify addentify addentify addentification addentify addentify adde | r (participate of the asset of | coants coants coants di l cons ked t ents applic that | an inf will s sent d o sign (s), in cable; will t | ocume or be format ) that v | onsen onsen ont with given tion s ( ( ( | t document de transfer de tran | ocumenne signature sent sent 4/24/24/24/24/24/24/24/24/24/24/24/24/24 | nent) t, but c nature any s sis stu dified 7/202- | ent) tatem dy. Th | ents ents se | of nev | provide<br>w | ed) | |
| 7. | Attacinfor any Nam Click Cons | Writt Altera Altera Altera Waive Waive Con HIP here ent f conne | en/sigr<br>tition of<br>er of sig<br>er of sig<br>er of co<br>er of co<br>pies of<br>on/find<br>at or pa | the elerconsent and info msent (p the inf ings or arental 27-202 orizatio in an IR abmitted section | ments of will be a primed consent of consent | consent (ints will not consent to addentify addentification addentification addentification addentify addentification addentification addentification addentification addentific | compliance on sent Terild compens | sign : coants d) I cons ked t ents applic that mnce)(I | an infi will s sent d o sign o sign (s), in cable) will t | ocume ocume or be format ) that v | nt with given tions so will be d. ( | t document de t document transcription de transcription d | wmen sign sent sent sent 4/2 4/2 eparii | nent) it, but contained any sample student any samp | esection ent) ttatem dy. Th | ents ents se | of nev | provide<br>w | ed) | |
| | Attachinfor any Nam Click Cons Pers - nor If the | Writt Altera Al | en/sigrition of other soft of significant of the soft of significant of the soft of significant of significant of significant or particular soft of significant of signific | the elerconsent med info msent (p the infi ings or mental 27-202 orizatio in an IR abmitted section incomp | ments of will be a participar of consense of the participar of the | consent (ints will not consent to addension document Consent to addension document Consent to addension document Consent to addension document Consent to addension document Consent Consent to addension document Consent Consent Consent to addension document Consent Conse | compliar consent, please | constants | an info | instruction in the control of the co | d consended to con | t document de t document transcription to the trans | ocumen he signature sent sent sent sent sent sent sent sen | any suits studified 7/202- | ent) tatem dy. Th 1 8:34 | ents ents se | of nev | provide<br>w | ed) | |
| .7. | Attachinfor any Nam Click Cons Pers - nor If the | Writt Altera Altera Waive Waive Ch commati asse Con HIP here ent f onne above cribe | en/sigrition of other soft of significant of the soft of significant of the soft of significant of significant of significant or particular soft of significant of signific | the elertonsent in the elerton sent (property of the infings or arental property or ization in an IR ibmitted section in compound in the incompound in the incompound in the important in the important | ments of will be a participar of consense of the consense of t | consent (ints will not consent to addension document Consent to addension document Consent to addension document Consent to addension document Consent to addension document Consent Consent to addension document Consent Consent Consent to addension document Consent Conse | compliar consent, please | constants | an info | instruction in the control of the co | d consended to con | t document de t document transcription to the trans | ocumen he signature sent sent sent sent sent sent sent sen | any suits studified 7/202- | ent) tatem dy. Th 1 8:34 | ents ents se | of nev | provide<br>w | ed) | |

| UP-21-00030 | - CO/ | D-19 and Preventive Health Behaviors | | 4/29/21, 8:48 AM |
|---|---|---|---|---|
| | | In a waiting room, open ward, group, or public setting | | |
| | ~ | Online, over the telephone, by mail, or via fax | | |
| | | Other | | |
| | | TE: When participants sign the informed consent electro<br>led to them. | nically, a copy of the informed consent document mus | be |
| 24.9. | | ribe how you will assess the individual's comprehen<br>ding understanding of the voluntary nature of partici | | te, |
| | ~ | An assessment tool will be used. (attach a copy of t | ne tool below) | |
| | | This will be verbally assessed. Individuals will be asked you being asked to do? (2) What question is this study t this study? (4) How often will you need to come in for st study and your standard medical care? (6) What should | ying to answer? (3) What are the potential risks of par<br>udy visits? (5) What is the difference between participa | ticipating in |
| | | Other (specify below) | | |
| | 24.9. | I. Assessment Tool: | | |
| | | Name Ver | sion Modified | |
| | | Quiz(0.02) 0.02 | 1/7/2021 3:06 PM | |
| 24.10. | | ribe all measures that will be taken during the recrui<br>uate time to consider participation and to safeguard<br>pply) | | |
| | <b>~</b> | The informed consent process will begin with a con most likely to assist a prospective participant in uno participate in the research | | |
| | ~ | They will not be forced, threatened or coerced in an or other form of constraint will be used to recruit incenrolled subjects. (Note: "Coercion" is the use or the influence" is when an individual who is in a position inappropriate or excessive manipulation to gain powersearch subject). "Constraint" means force, obligations or the constraint of the cons | lividuals to participate in this research or to retain<br>reat of the use of force to gain compliance. "Undue<br>of authority (e.g., physician, teacher, employer) ex<br>rer and compliance over a vulnerable individual (po | currently<br>e<br>erts |
| | ~ | They will not be punished or denied something which health services to which an individual would otherw research or choose to withdraw early from participa | ise be entitled) if they choose not to participate in t | |
| | ~ | They will be given an adequate amount of time to co study procedures. | nsider participation in the study relative to the initi | ation of |
| | ~ | The information presented to individuals during rec<br>informed consent document/informed consent scrip | | е |
| | ~ | The recruitment and consent process will not promi<br>in the informed consent document/informed consen | | is outlined |
| | ~ | The recruitment and consent process will take place confidentiality. | in an area in which it is possible to maintain priva | cy and |
| | | They will be given the opportunity to take the informed of family, friends and/or others before making a definitive of | | n with their |
| | | They will receive payment for their participation, but the (not an inducement for participation), and receipt of the the study. (Note: The specific method, schedule, and an | payment will not be contingent upon the individual's co | mpletion of |
| https://istar.u | sc.edu | istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.h | tml | |

| | application.) |
|---|---|
| | Other (explain below) |
| 8 19 | Financial Obligation and Compensation |
| .1. | Financial Obligation: Choose the response that best describes the cost to participants. |
| | All costs are covered by the sponsor or funder. |
| | Research costs are paid by the sponsor or funding agency; routine health care costs are the responsibility of the participants and/or their healthcare plans. |
| | All costs are the responsibility of the participants and/or their healthcare plans. |
| | O Drug trials sponsored by the National Cancer Institute or other national institutes. |
| | There are no costs related to participation. |
| | Other |
| .2. | Payment for Participation: Describe how much, if any, financial or other form of compensation will be provided to the subject/family. Describe the requisite conditions that must be fulfilled to receive full or partial compensation. Describe the proposed method of timing and disbursement. If children are involved, please specifically address how the compensation will be distributed to children. Individuals who consent to the study and complete the baseline survey will receive a \$5 gift card. They will also be eligible for a raffle. We will raffle off 20 gift cards at \$250 per card. We also have financial incentives for vaccine take-up. Specifically, we will randomly vary incentives for vaccination at \$10 and \$50. These incentive values are in line with the prior literature. For example, Bronchetti, Huffman, and Magenheim (2015) paid college students \$30 for flu vaccinations in 2012. In addition, the \$50 incentive is in-line with 2 hours of time at the minimum |
| | wage plus transportation costs. As noted in our protocol, many behavioral economic studies that have been approved by IRBs at peer institutions vary incentive amounts for the same activitiy. |
| | This design will enable CCHS to understand the potential costs and benefits of a financial assistance program to increase vaccinations more generally, e.g., influenza vaccination, something they are considering for vaccinations generally, i.e., not only COVID-19 vaccination. Without varying these incentives, we cannot provide CCHS with a good estimate of how to cost-effectively design such a program in the future. While we understand concerns about equity, deception, which has been suggested by the IRB as a way to equalize payments ex-post, is not viewed as acceptable practice in our field (economics). In addition, we think it would be potentially harmful to use deception to study infectious disease in low-income disparity populations. |
| 5. | Participant Privacy and Data Confidentiality |
| .1. | <b>Privacy Protections</b> : Privacy is a participant's ability to control how other people see, touch, or obtain information about his/her self. Violations of privacy can involve circumstances such as being photographed or videotaped without consent, being asked personal questions in a public setting, being seen without clothing, being observed while conducting personal behavior, or disclosing information about abortions, HIV status, or illegal drug use. |
| | Select the provisions to protect the privacy of the individual during screening, consenting, and conduct of the research: (check ALL that apply) |

| | | Data \ | will be captured and reviewed in a private setting. |
|---|---|---|---|
| | | Only a | authorized research study personnel will be present during research related activities. |
| | ~ | The c<br>resea | ollection of information about participants is limited to the amount necessary to achieve aims of the rch. |
| | | | ipants will not be approached in a setting or location that may constitute an invasion of privacy or could potentially atize them. |
| | | Other | (specify below) |
| <u>2</u> . | unde | erstandi | <b>ality Precautions</b> : Confidentiality is an extension of the concept of privacy; it refers to the participant's ng of, and agreement to, the ways identifiable information will be collected, stored, and shared. Identifiable can be printed information, electronic information, or visual information such as photographs. |
| | How | will th | e research data/specimens be labeled? (check ALL that apply) |
| | | Data a | and/or specimens will be directly labeled with personal identifying information. (Identifiable) |
| | ~ | | and/or specimens will be labeled with a code that the research team can link to personal identifying nation. (Coded) |
| | | | and/or specimens will not be labeled with any personal identifying information, nor with a code that the research can link to personal identifying information. (Anonymous) |
| | | Other | (explain below) |
| | Ctua | | |
| 3. | Stud | ly data | /specimen will be stored: |
| 3. | Stud | | /specimen will be stored: |
| 3. | Stud | <b>ly dat</b> a | /specimen will be stored: |
| 3. | | ly data<br>Physic | /specimen will be stored: |
| 3. | | ly data<br>Physic | /specimen will be stored: cally conically |
| ١. | | ly data<br>Physic | /specimen will be stored: cally ronically ch devices will have study data: |
| ı. | | ly data<br>Physic | /specimen will be stored: cally ronically ch devices will have study data: Local computers/laptops |
| 3. | | ly data<br>Physic | Aspecimen will be stored: cally ronically ch devices will have study data: Local computers/laptops Removable drives (USB, external drives) |
| 3. | | ly data<br>Physic | Aspecimen will be stored: cally ronically ch devices will have study data: Local computers/laptops Removable drives (USB, external drives) Local Server(s) |
| i. | | ly data<br>Physic | Aspecimen will be stored: cally conically ch devices will have study data: Local computers/laptops Removable drives (USB, external drives) Local Server(s) External Servers (including cloud based services) Which company/organization will be providing the service? |
| 3. | | Physic Electr White | Ispecimen will be stored: cally ronically ch devices will have study data: Local computers/laptops Removable drives (USB, external drives) Local Server(s) External Servers (including cloud based services) Which company/organization will be providing the service? Box.com Note: Please ensure that the third party♠s technical infrastructure meets or exceeds the minimum |


| | | ~ | Electronic data will be stored with appropriate electronic safeguards, such as unique usernames/passwords, and limited to authorized study personnel. Dual factor authentication will be used, if feasible. |
|---|---|---|---|
| | | | Copying and use of study related materials will be restricted |
| | | ~ | Security software (firewall, antivirus, anti-intrusion) will be installed and regularly updated in all servers, workstations, laptops, and other devices used in the study |
| | | ~ | All computers with access to study data will be scanned regularly (for viruses and spyware, etc.) and problems will be resolved |
| | | | Data stored on a removable drive will be encrypted and have proper access controls |
| | | ~ | Data transfer will be encrypted |
| 6.4. | ager | | ied data and/or specimens be sent outside the institution to a third party (such as a study sponsor, federal another institution)? No |
| 6.5. | Wha | t will h | appen to the research data and/or specimens at the conclusion of the study? (check ALL that apply) |
| | <b>~</b> | data/s | t identifiers and/or the key to the codes will be destroyed upon completion of the research (all specimens will be stripped of identifying information and/or the key to codes destroyed, paper documents ded, electronic files purged, electronic media securely erased) |
| | | Retair | ned for study record keeping purposes per institutional policy |
| | | Retaii | ned by the investigator for future research use |
| | | Retair | ned for future research use (submit data or tissue to an existing repository/bank) |
| | | Restri | cted use data will be destroyed or returned to the source |
| | | | ect or indirect identifiers are being collected. The anonymous data and/or specimens will be retained at the tion of the investigator |
| | | | esearch is a clinical trial conducted under FDA regulations. Direct identifiers and/or the key to the codes will be<br>byed as directed by the sponsor (IND/IDE holder) in accordance with FDA regulations |
| | | The N | IIH requires that the records be retained for three years following the completion of the study |
| | | Other | (specify below) |
| 6.6. | - | 59 S 57 | ve, or plan to apply for, a Certificate of Confidentiality for this study? No |
| | NOT | E: NIH | -funded research in which identifiable, sensitive information is used, including research that: |
| | | | ts the definition of human subjects' research, including exempt research in which subjects can be |
| | 1 | ls co | tified<br>Illecting or using human bio specimens that are identifiable or that have a risk of being identifiable<br>Ives the generation of individual level human genomic data<br>Ives any other information that might identify a person |
| | is au | | cally protected by a certificate of confidentiality from the NIH |

# 27. Risk/Benefit Assessment - Risks

| | | s, Discomforts and Potential Harms: Describe the risks associated with each research intervention. Include ideration of physical, psychological, social, and other factors. (check all that apply) |
|---|---|---|
| | | Discrimination based on genetic findings. |
| | | Some people may find it upsetting to learn that they have certain mutations or errors in genes that could lead to future health problems for themselves or their children. |
| | ~ | Some of the questions may make the participant feel uneasy or embarrassed. |
| | ~ | There is a small risk that people who are not connected with this study will learn a participant sidentity or their personal information. |
| | | The participants are providing highly sensitive, personal information in this study. If people not connected with the study learn this information, they could have problems getting a new job, keeping their current job, finding housing, or getting insurance (health, disability, or life insurance). In highly unlikely situations, they could be charged with a crime. |
| | | Biomedical risks, including drug, device, biologics, radiation, surgery or other research procedures (please specify). |
| | | The research includes the risk or disclosure that a participant may engage in self-harm or attempt suicide. |
| | | Venipuncture risks including: mild discomfort (or pain), bruising and swelling around the puncture site, dizziness or fainting, or infection (rare). |
| | | Other (specify below) |
| .2. | Desc | ribe the precautions that will be taken to minimize risks/harms. (check all that apply) |
| | ~ | We will use our best efforts to keep the findings in this study as confidential as possible. |
| | ~ | Subjects can choose to skip or stop answering any questions that make them uncomfortable. |
| | <b>~</b> | Data will be coded and identity stored separate from data. |
| | | Data will be collected anonymously. |
| | | Data will be collected anonymously. Biomedical precautions, including precautions relating to drugs, devices, biologics, radiation, surgery or other research procedures (please specify). |
| | | Biomedical precautions, including precautions relating to drugs, devices, biologics, radiation, surgery or other research |
| | | Biomedical precautions, including precautions relating to drugs, devices, biologics, radiation, surgery or other research procedures (please specify). |
| 28. | Ris | Biomedical precautions, including precautions relating to drugs, devices, biologics, radiation, surgery or other research procedures (please specify). Venipuncture by individuals certified and privileged to perform the procedure. |
| 28.<br>8.1. | | Biomedical precautions, including precautions relating to drugs, devices, biologics, radiation, surgery or other research procedures (please specify). Venipuncture by individuals certified and privileged to perform the procedure. Other (specify below) |
| | | Biomedical precautions, including precautions relating to drugs, devices, biologics, radiation, surgery or other research procedures (please specify). Venipuncture by individuals certified and privileged to perform the procedure. Other (specify below) k/Benefit Analysis - Potential Benefits and Alternatives |

| 21-0003 | 30 - CO\ | /ID-19 and Preventive Health Behaviors | 4/29/21, 8:48 / |
|---|---|---|---|
| | | Improvement in some or all of participants' surviv | al or longevity |
| | | Information gained from testing or monitoring pro | pedures |
| | | Provision of drug or device | |
| | | Reduced side effects | |
| | | Other (explain below) | |
| 28.2. | Descr | ibe potential benefits to society, if any. (check | all that apply) |
| | | The advancement of knowledge | |
| | | A new treatment or therapy for the condition unde | r study |
| | | None | |
| | ~ | Other (explain below) | |
| | 28.2.1 | Describe other potential benefits to society If we can increase vaccine take-up, we increa evidence on how to increase vaccine take-up | se the likelihood of herd immunity. We will also generate broader |
| 28.3. | What | are the alternatives to participation? (check al | that apply) |
| | ~ | Not participating | |
| | | Continue current medical care for their condition | |
| | | Participation in other research studies | |
| | | Palliative care | |
| | | No treatment or therapy | |
| | | Participate in other subject pool activities | |
| | | Other (specify below) | |
| 28.4. | Risks | in relation to benefits: | |
| | | The potential benefits to the research participants | justify exposure of the participants to the risks. |
| | ~ | The potential benefits to humanity justify exp | osure of the participants to the risks. |
| | | Other (specify below) | |
| 35 | Ic th | ne HIPAA Privacy Rule Appl | icable? |
| JJ. | io (I | ic iminati iivacy naic appi | IOUDIC. |


| | <ul> <li>Look at clinic logs to identify potential research participants</li> </ul> | |
|---|---|---|
| | <ul> <li>Record demographic information obtained from medical records (paper or electronic)</li> </ul> | |
| | Record health information obtained from medical records (paper or electronic) Obtain information obtained from medical records (paper or electronic) | |
| | <ul> <li>Obtain information from laboratory reports, pathology reports, radiology reports or images, or other reports from<br/>medical or mental health testing and treatment</li> </ul> | |
| | Obtain information from medical billing records | |
| | Record or use medical record numbers or other information that could be used to identify an individual (review the | list |
| | of HIPAA identifiers below) | liot |
| | Name/Initials | |
| | <ul> <li>Street address, city*, county*, precinct*, zip code*, or equivalent geocodes*</li> </ul> | |
| | <ul> <li>All elements of dates (except year) directly related to an individual (date of birth, admission date, discharge</li> </ul> | |
| | date, date of death)* | |
| | <ul> <li>Elements of date, including year, for persons 90 or older</li> </ul> | |
| | Telephone number | |
| | • Fax number | |
| | Electronic mail address | |
| | Social Security Number | |
| | Medical record number | |
| | <ul> <li>Health plan identification number</li> <li>Account number</li> </ul> | |
| | Certificate/license number | |
| | Vehicle identifiers and serial numbers, including license plate number | |
| | Vertice identifiers and serial number Device identifiers and serial number | |
| | Web addresses (URLs): Internet IP addresses | |
| | <ul> <li>Biometric identifiers, including finger and voice print</li> </ul> | |
| | <ul> <li>Full face photographic images and any comparable images</li> </ul> | |
| | <ul> <li>Any other unique identifying number, characteristic, or code*</li> </ul> | |
| | ■ Yes No | |
| 35.2. | 2. Do you intend to record data that contains any of the 18 elements defined by HIPAA as identifiers (listed above), | in |
| | your research? | |
| | ■ Yes ○ No | |
| 35.3. | <ol><li>Are you going to record only the personal identifiers marked with an asterisk (*)? If so, you may be able to obtain</li></ol> | |
| | use such health information from a healthcare provider for research purposes without an authorization. Under the | |
| | HIPAA Privacy Rule, this data constitutes a elimited data sete. if you are creating or obtaining a limited data se | et, you |
| | must complete a Data Use Agreement. Attach a copy of the signed Data Use Agreement below. | |
| | Name Version Modified | |
| | There are no items to display | |
| | There are no terms to display | |
| 35.4. | 4. Will you be recording HIV data? | |
| 5.54 10 | Yes No | |
| | les and | |
| 35.5. | 5. Will you be collecting or accessing mental health records from a mental health practitioner? | |
| | Yes No | |
| 35.6. | 6. Will you be collecting or accessing substance abuse treatment records? | |
| | Yes No | |
| | USC Template Data Use Agreement | |
| | ** If your Data Use Agreement does not use USC�s template form, please contact USC�s Office of Compliance at | |
| | complian@usc.edu or 213-740-8258 to submit the Data Use Agreement for further review and approval. | |

• Look at medical records (paper or electronic) to identify potential research participants

## 36. HIPAA Analysis

https://istar.usc.edu/istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.html


This screen is only required if you indicated HIPAA is applicable by answering "yes" to Question 35.1. If you are using or accessing protected health information in order to identify potential participants, indicate if you will be applying for a Partial Waiver of HIPAA Authorization for the purposes of screening and recruiting Partial Waiver of HIPAA Authorization for screening, recruiting, and identifying participants None of the Above 36.2. If you are using or accessing protected health information to conduct the research, please select whether you will be obtaining authorization from the participant or requesting a Full Waiver of HIPAA Authorization. Obtaining HIPAA authorization from participant Full Waiver of HIPAA Authorization ( ) Both Click here to download the "Instructions for Completing HIPAA Research Authorization Form" and the HIPAA research authorization forms approved by the USC Office of Compliance (scroll down to "Research (300))". I agree to use the current HIPAA research authorization forms and make only those changes described in the Instructions for Completing HIPAA Authorization Form. I modified the HIPAA research authorization form and received approval from the USC Office of Compliance to 38. Partial Waiver of HIPAA Authorization This screen is required only if HIPAA is applicable and you indicated you are requesting a Partial Waiver of HIPAA Authorization (Question 36.1.) If you are applying for a partial waiver of authorization for the purposes of screening, recruitment, and subject identification, provide justification per 45 CFR 164. 38.1. How will you protect PHI/ePHI (Protected Health Information) from improper use and disclosure? (check all that apply) PHI/ePHI will be used only for the purposes of assessing eligibility and identifying potential participants. All source and research documents containing PHI/ePHI will be stored and maintained in a locked/password protected area accessible only to study staff. Study data will be coded or de-identified prior to being sent outside the study team. Other 38.2. How will you destroy identifiers at the earliest opportunity consistent with the conduct of the research? (check all that No identifiers or links to identifiers will be recorded during the data collection process.

Direct or Coded Identifiers will be maintained only until the study is completed. After that, the identifiers will be

https://istar.usc.edu/istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.html

shredded and electronic records purged.


| IJ | P. | 21- | -00 | 003 | ) - | COVID | -19 ar | d Preve | entive | Health | Behav | riors |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

4/29/21, 8:48 AM

| | The link between study participants and study ID numbers will be destroyed (shredded/purged) when study activities are complete. |
|---|---|
| | Other |
| 38.3. | By checking the "I Agree" box you are providing assurance that PHI/ePHI will not be reused or disclosed to any other person or entity except (a) as required by law, (b) for authorized oversight of the research study, or (c) for other research for which the use or disclosure of the PHI/ePHI is permitted by the Privacy Rule. |
| | ✓ I Agree |
| 38.4. | The research could not practicably be conducted without the requested waiver or alteration because: (check all that apply) |
| | PHI/ePHI is required to identify potential participants who meet the eligibility criteria. |
| | Other |
| 38.5. | The research could not practicably be conducted without access to and use of the PHI/ePHI because: (check all that apply) |
| | PHI/ePHI is required to identify potential participants who meet the eligibility criteria. |
| | During the recruitment process, PHI/ePHI is needed in order to contact potential participants. |
| | ☐ Other |
| 38.6. | By checking the "I Agree" box you are providing assurance that PHI/ePHI requested will be the minimum amount necessary to conduct the research or meet the research objectives. |
| | ✓ I Agree |

## 39. Conflict of Interest Information

39.1. Indicate the Study team member(s) that have a potential conflict of interest. For each person to be designated, click on his/her name and select the disclosure(s) that should be associated with this study.

| Study Staff | Role | COI Annual Disclosure Status | Conflicts |
|---|---|---|---|
| Mireille Jacobson | Principal Investigator | Current: due on 7/31/2021 | No conflicts identified |
| Tom Chang | Co-Investigator | Current: due on 7/31/2021 | No conflicts identified |

## 40. Additional Supporting Documents

40.1. Attach any other documents that have not been specifically requested in previous questions, but are needed for IRB review.

| Name | Version Modified | |
|---|---|---|
| MIT JPAL - SMART IRB Determination(0.01) | 0.01 | 3/22/2021 11:54 AM |
| NBER IAA(0.01) | 0.01 | 4/28/2021 8:50 AM |

https://istar.usc.edu/istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.html


40.2. If there is any additional information that you wish to communicate about the study include it below. Please note, this section should not be used instead of the standard application items.

As mentioned elsewhere, many behavioral economics studies vary incentives for the same behavior. The amended protocol lists several recent studies that are relevant. Here we list a few others for the IRB's consideration:

1) Volpp, K.G., Loewenstein, G., Troxel, A.B. et al. A test of financial incentives to improve warfarin adherence. BMC Health Serv Res 8, 272 (2008). https://doi.org/10.1186/1472-6963-8-272. https://bmchealthservres.biomedcentral.com/articles/10.1186/1472-6963-8-272

Study participants were randomized to be entered into a daily lottery of \$10 or \$100 for warfarin adherence.

This study was approved by the IRB at University of Pennsylvania.

2) Alicea Lieberman, Ayelet Gneezy, Emily Berry, Stacie Miller, Mark Koch, Chul Ahn, Bijal A. Balasubramanian, Keith E. Argenbright and Samir Gupta, Financial Incentives to Promote Colorectal Cancer Screening: A Longitudinal Randomized Control Trial Cancer Epidemiol Biomarkers Prev November 1 2019 (28) (11) 1902-1908; DOI: 10.1158/1055-9965.EPI-19-

Patients were randomized to receive outreach alone or outreach and either incentives of \$5 or \$10 for completion of a fecal immunochemical test (FIT).

This study was approved by the IRB at Texas Southwestern Medical Center

3) Beshears, John, Hae Nim Lee, Katherine L. Milkman, Robert Mislavsky, and Jessica Wisdom, Creating Exercise Habits Using Incentives: The Tradeoff between Flexibility and Routinization, Management Science https://pubsonline.informs.org/doi/10.1287/mnsc.2020.3706

This study tried to increase exercise. Participants were randomly assigned to a control that received daily reminders, daily reminders and either \$3 or \$7 for each gym visit in a 4-week period or daily reminders and either \$3 or \$7 for each gym visit within a 2-hour pre-selected window in a 4-week period.

This study was approved by the IRBs at Harvard, the National Bureau of Economic Research and the University of Pennsylvania.

#### 41. Feasibility Information for Scientific Review

This page is required when the research has not yet undergone scientific review.

41.1. What is the expected duration of the accrual period?

1 month for baseline study recruitment

- 41.2. Describe any competing studies at USC (i.e. studies with similar inclusion/exclusion criteria and similar recruitment timeframes). Include investigator names and study titles, if known.
  None that I am aware of.
- 41.3. Describe the study team's expertise and experience relevant to this study.

The study investigators have been collaborating with CCHS on an internally-funded project, Behavioral Response to COVID-19 Testing, inc May 2020. In that work, we are fielding an initial and follow-up survey to Medicaid managed care enrollees coming to CCHS for clinician-ordered blood lab work as well as to individuals coming to county public health diagnostic testing sites. A subset of the blood lab sample is randomly offered free COVID-19 antibody testing, with the goal of understanding how antibody testing affects behaviors. We ceased recruiting at the end of the week of September 14. Since July, about 2,100 respondents have filled out an initial survey and nearly 1,800 have been invited via text and/or email to a follow-up survey. At present, we have just over 1330 follow-up surveys of these individuals via email or text to the follow-up surveys completed. Despite offering only a \$5 incentive for survey completion and the chance to win a \$500 gift card, the follow-up survey response rate has remained at about 74% for the past month. That work effectively serves as a pilot for this

https://istar.usc.edu/istar/sd/Doc/0/JGAV60L8DC8UMQC1TH8OULIG00/fromString.html

project.

41.4. Describe the resources required to conduct this study and plans for accessing them. Examples of resources include equipment, facilities, and materials.

| | | will use the USC RedCAP system. We have funds to hire a research manager and<br>work. | d a research assistant to help implement | |
|---|---|---|---|---|
| 42. | Cli | nical Data Warehouse | | |
| This s | creen | is required if you indicated the use of a clinical data warehouse in 13.3.1 or 24.1 | | _ |
| 42.1. | Whi | ch Clinical Data Warehouse(s) will you be using? | | |
| | | Keck Medicine of USC | | |
| | | LA County/DHS | | |
| | ~ | Other | | |
| | 42. | Please Specify the other clinical data warehouse(s) you will be using: Contra Costa Health Services Data Warehouse | | |
| 42.2. | Whi | ch of the following HIPAA Identifiers will you be recording? | | |
| | ~ | Name | i | |
| | ~ | Address | | |
| | | All elements (except years) of dates related to an individual | | |
| | <b>~</b> | Telephone numbers | | |
| | | Fax number | | |
| | ~ | Email address | | |
| | | Social Security Number | | |
| | ~ | Medical record number | | |
| | | Web Universal Resource Locators (URLs) | | |
| | | Device identifiers and serial numbers | | |
| | | Vehicle identifiers and serial numbers, including license plate numbers | | |
| | | Internet Protocol (IP) addresses | | |
| | | Biometric identifiers, including finger and voice prints | | |
| | | Health plan beneficiary numbers | | |

https://istar.usc.edu/istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.html

| UP-21-0003 | 0 - COVID-19 and Preventive Health Behaviors | 4/29/21, 8:48 AM |
|---|---|---|
| | Full-face photographs and any comparable images | |
| | Account numbers | |
| | Any other unique identifying number, characteristic, or code | |
| | Certificate/license numbers | |
| | None of the 18 HIPAA identifiers will be recorded or stored as part of this study. | |
| 42.3. | Do you intend to contact people identified from the data obtained from the clinical data warehouse? Yes No | |
| | 42.3.1. Please indicate how you will be contacting them: E-mail or text. | |
| 99 | Instructions for Submission | |
| You ha | ave reached the end of the application. When you are sure of the content, the following steps may be taken to spplication for review. | <br>submit |
| 2.<br>3.<br>4.<br>5. | Click the <b>"Finish"</b> button on the top or bottom application navigator bar to return to the workspace. Use the <b>Hide/Show Errors</b> above to determine that all sections of the application are filled out correctly. Use the <b>"Send Study Ready Notification"</b> activity to send an email to the Principal Investigator and Co-Investigators instructions for reviewing and submitting the application. <b>All listed Co-Investigators (indicated in item 2.1.) must use the "Agree to Participate" activity and answer yes.</b> Once all the Co-Investigators have agreed to participate, the <b>Principal Investigator</b> (indicated in item 2.1.) can submit application by using the <b>"Submit Application to"</b> , where indicates the IRB you are submitting to. The PI will have to check the PI endorsement box. The PI will also have to check the student endorsement box if it is a The application is submitted. The state indicator in the top left of the workspace will no longer display Pre Submission. The PI and Study Contact Person will receive an email confirming the application has been submitted. | the |
| 4.4. F | unding Source | |
| Please | enter the fields below and click 'OK' when done. | |
| 4.4.1. | * Name of Sponsor:<br>National Institutes on Aging | |
| 4.4.2. | * Named Principal Investigator:<br>Joe Doyle and David Laibson | |
| 4.4.3. | Institution awarded the grant-award:<br>National Bureau of Economic Research | |
| 4.4.4. | Grant-award number provided by the Sponsor: 5P30AG034532-12 | |
| 4.4.5. | Title of the Funding Project, if applicable: | |
| 4.4.6. | * Type of Funding: Federal: Program Project/Multiple Project Grant * | |
| https://istar. | usc.edu/istar/sd/Doc/0/JGAV60L8DC8UMQC1TH8OULIG00/fromString.html | |

4.4.7. Attach a copy of the proposal/contract/grant with the project budget. Copies of the documents submitted to the funding agency, including the budget detail, should be submitted. (salary information need not be displayed or included.)

Name Version Modified

There are no items to display

| 6d.1 C | ther Site | |
|---|---|---|
| Please | complete the | form below and click 'OK' when done. |
| 6d.1.1. | * Site Name:<br>Contra Costa | :<br>a Health Services |
| 6d.1.2. | * Address:<br>333 C Street | , Martinez, CA 94553 |
| | ☐ Internat | tional (Check here if [site] is not in the United States) |
| 6d.1.3. | | escribe the activities that will occur at [site]: ruiting from members of CCHS,. |
| 6d.1.4. | Determinir | ng Engagement: |
| | Will [site] ۽ | personnel conduct any of the following activities? |
| | * 6d.1.4.1. | Recruitment and Consent: |
| | | Inform potential participants of the availability of the research, provide study contact information, or seek permission for investigators to contact the potential participants? Yes No |
| | | Obtain informed consent from the research participants? Yes No |
| | * 6d.1.4.2. | Participant Data and Information: |
| | | Release to the study investigators data or information about the research participants that have been collected for non-research purposes? Yes No |
| | | Obtain identifiable data or information about the research participants solely for the purposes of the research project? Yes No |
| | * 6d.1.4.3. | Participant Contact and Intervention: |
| | | Interact with the research participants for routine care, follow up or commercial services? Yes \int No |
| | | Interact or intervene with research participants for research purposes (including performing procedures or manipulating the environment)? Yes No |

https://istar.usc.edu/istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.html


| | | D-19 and Preventive Health Behaviors | | | |
|---|---|---|---|---|---|
| * 6d.1.5. | - | [site] receive any direct federa | al support for th | s research? | |
| Vauron | | Contractor | in the receased | Veu must answer the fellow | din at |
| your an | swers | indicate that [site] is engaged | in the research. | You must answer the follow | ving. |
| 40. | | List IDD Andrews | | | |
| 1.8. l | _ | which IRB Authorization Agree MART IRB | ement will [Site] | rely on the USC/CHLA IRB to | o review this study? |
| | • 0 | ther | | | |
| | | e the name of the agreement: | | | |
| | | d the agreement, if available: | | | |
| | 5 | <del></del> ∞ | | | |
| 6d.1.9. | Plea: | se attach a letter from [site] acl<br>e | | t the study may be conduct<br>on Modified | ed there. |
| | 周 | CCHS IRB memo.pdf(0.01) | 0.01 | 3/15/2021 6:20 PM | |
| | _ | | | | |
| 6d.1.9. | | | | | g consent or conducting study<br>Yes |
| | Will a | any of the personnel at [site] ca<br>edures? (Deprecated Field - use<br>s, indicate under which categor<br>below. (Deprecated Field - old 6 | arry out researced to be 6c.1.3 o | n activities such as obtainin only used for old studies) | |
| | Will a | any of the personnel at [site] ca<br>edures? (Deprecated Field - use<br>s, indicate under which categor<br> below. (Deprecated Field - old 6<br> Short Description | arry out researced to be 6c.1.3 or<br>ry(ies) [site] is e<br>6c.1.4 only use | n activities such as obtaining only used for old studies) ngaged (see guidance) and a for old studies) | Yes No ttach a copy of the IRB approval from |
| | Will a | any of the personnel at [site] ca<br>edures? (Deprecated Field - use<br>s, indicate under which categor<br> below. (Deprecated Field - old 6<br> Short Description | arry out researced to be 6c.1.3 or ry(ies) [site] is e 6c.1.4 only usedward through a gi | n activities such as obtaining only used for old studies) ngaged (see guidance) and a for old studies) | Yes No |
| | Will a | any of the personnel at [site] caedures? (Deprecated Field - uses, indicate under which category below. (Deprecated Field - old 6 Short Description (1) Institutions that receive an avexempt human subjects research | arry out researced to be 6c.1.3 or only used ward through a gradu. | n activities such as obtaining only used for old studies) ngaged (see guidance) and a differ old studies) ant, contract, or cooperative a | Yes No ttach a copy of the IRB approval from |
| | Will a | any of the personnel at [site] caedures? (Deprecated Field - uses, indicate under which category below. (Deprecated Field - old 6 Short Description (1) Institutions that receive an avexempt human subjects research (2) Institutions whose employee performing invasive or noninvas | arry out researced to be 6c.1.3 or only used ward through a graph. | n activities such as obtaining only used for old studies) ngaged (see guidance) and a differ old studies) ant, contract, or cooperative a guidance or research purposes with | Yes O No |
| 6d.1.9. | Will a | any of the personnel at [site] caedures? (Deprecated Field - uses, indicate under which category below. (Deprecated Field - old 6 Short Description (1) Institutions that receive an avexempt human subjects research (2) Institutions whose employee performing invasive or noninvas (3) Institutions whose employee manipulating the environment. | arry out researce and to be 6c.1.3 or only used ward through a grade. s or agents intervive procedures. | n activities such as obtaining only used for old studies) ngaged (see guidance) and a differ old studies) ant, contract, or cooperative a ene for research purposes with | Yes No |
| | Will: proc | any of the personnel at [site] caedures? (Deprecated Field - uses, indicate under which category below. (Deprecated Field - old 6 Short Description (1) Institutions that receive an avexempt human subjects research (2) Institutions whose employee performing invasive or noninvas (3) Institutions whose employee manipulating the environment. | arry out researce and to be 6c.1.3 or only used ward through a grade. sor agents intervive procedures. sor agents intervive procedures. | n activities such as obtaining only used for old studies) on gaged (see guidance) and a differ old studies) ant, contract, or cooperative a gene for research purposes with ct for research purposes with | Yes No |
| | Will: proc | any of the personnel at [site] caedures? (Deprecated Field - uses, indicate under which category below. (Deprecated Field - old 6 Short Description (1) Institutions that receive an avexempt human subjects research (2) Institutions whose employee performing invasive or noninvas (3) Institutions whose employee manipulating the environment. (4) Institutions whose employee (5) Institutions whose employee | arry out researce of to be 6c.1.3 or ry(ies) [site] is e 6c.1.4 only use ward through a gish. s or agents intervive procedures. s or agents intervive s or agents intervive s or agents obtains or agents obtains or agents obtains | n activities such as obtaining only used for old studies) ngaged (see guidance) and a differ old studies) ant, contract, or cooperative a sene for research purposes with the informed consent of human for research purposes identifications. | Yes No |
| 6d.1.10. | Will i | any of the personnel at [site] caedures? (Deprecated Field - uses, indicate under which category below. (Deprecated Field - old 6 Short Description (1) Institutions that receive an avexempt human subjects research (2) Institutions whose employee performing invasive or noninvasive or noninv | arry out researce of to be 6c.1.3 or ry(ies) [site] is e 6c.1.4 only use ward through a gish. s or agents intervive procedures. s or agents intervive s or agents intervive s or agents obtains or agents obtains or agents obtains | n activities such as obtaining only used for old studies) ngaged (see guidance) and a differ old studies) ant, contract, or cooperative a sene for research purposes with the informed consent of human for research purposes identifications. | Yes No Ittach a copy of the IRB approval from Ingreement directly from HHS for the non- Ith any human subjects of the research by Ith any human subject of the research by any human subject of the research. |
| 6d.1.10.<br>6d.1 O | Will is process for year [site] | any of the personnel at [site] caedures? (Deprecated Field - uses, indicate under which category below. (Deprecated Field - old 6 Short Description (1) Institutions that receive an avexempt human subjects research (2) Institutions whose employee performing invasive or noninvasive or noninv | arry out researce and to be 6c.1.3 or only used ward through a grade. sor agents intervive procedures. sor agents intervive agents intervive procedures. sor agents obtains or agents obtains ource for the research | n activities such as obtaining only used for old studies) ngaged (see guidance) and a differ old studies) ant, contract, or cooperative a sene for research purposes with the informed consent of human for research purposes identifications. | Yes No Ittach a copy of the IRB approval from Ingreement directly from HHS for the non- Ith any human subjects of the research by Ith any human subject of the research by any human subject of the research. |

**6d.1.2.** \* Address: 400 Main Street E19-201 Cambridge, MA 02142 USA


| JP-21-00030 - | COVID-19 and | Preventive Health Behaviors | 4/29/21, 8:48 AM |
|---|---|---|---|
| | ☐ Internat | ional (Check here if [site] is not in the United States) | |
| 6d.1.3. | MIT/J-PAL i | scribe the activities that will occur at [site]:<br>s the funder. J-PAL gets their funding from foundations as well as donations. As such, this is technically<br>so they need IRB approval. | 'a sub- |
| 6d.1.4. | Determinin | g Engagement: | |
| | Will [site] p | ersonnel conduct any of the following activities? | |
| | * 6d.1.4.1. | Recruitment and Consent: | |
| | | Inform potential participants of the availability of the research, provide study contact informatic seek permission for investigators to contact the potential participants? Yes No | on, or |
| | | Obtain informed consent from the research participants? Yes No | |
| | * 6d.1.4.2. | Participant Data and Information: | |
| | | Release to the study investigators data or information about the research participants that have collected for non-research purposes? Yes No | e been |
| | | Obtain identifiable data or information about the research participants solely for the purposes research project? Yes No | of the |
| | * 6d.1.4.3. | Participant Contact and Intervention: | |
| | | Interact with the research participants for routine care, follow up or commercial services? Yes No | |
| | | Interact or intervene with research participants for research purposes (including performing pror manipulating the environment)? $\bigcirc \ \text{Yes} \ \bigcirc \ \text{No}$ | ocedures |
| * 6d.1.5. | Will [site] r | eceive any direct federal support for this research? No | |
| Your ans | wers indicat | te that [site] is engaged in the research. You must answer the following: | |
| 6d.1.8. U | Inder which I | RB Authorization Agreement will [site] rely on the USC/CHLA IRB to review this study? | |
| | Other | RB | |
| 6d.1.9. | Will any of t | he personnel at [site] carry out research activities such as obtaining consent or conducting stud | dy |
| ittps://istar.us | c.edu/istar/sd/D | oc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.html | |

| UP-21-00030 | 2 - COVID-19 and Preventive Health Behaviors 4/29/3 | 21, 8:48 |
|---|---|---|
| | procedures? (Deprecated Field - used to be 6c.1.3 only used for old studies) Yes No | |
| 6d.1.10. | If yes, indicate under which category(ies) [site] is engaged (see guidance) and attach a copy of the IRB approval (site] below. (Deprecated Field - old 6c.1.4 only used for old studies) | from |
| | Short Description | |
| | (1) Institutions that receive an award through a grant, contract, or cooperative agreement directly from HHS for the exempt human subjects research. | non- |
| | (2) Institutions whose employees or agents intervene for research purposes with any human subjects of the research performing invasive or noninvasive procedures. | ch by |
| | (3) Institutions whose employees or agents intervene for research purposes with any human subject of the research manipulating the environment. | h by |
| | (4) Institutions whose employees or agents interact for research purposes with any human subject of the research. | |
| | (5) Institutions whose employees or agents obtain the informed consent of human subjects for the research. | |
| | (6) Institutions whose employees or agents obtain for research purposes identifiable private information or identifiable biological specimens from any source for the research. | ole |
| 6d.1 O | Other Site | |
| Please o | complete the form below and click 'OK' when done. | |
| 6d.1.1. | * Site Name:<br>National Bureau of Economic Research (NBER) | |
| 6d.1.2. | * Address: | |
| | 1050 Massachusetts Ave, Cambridge, MA 02138 | |
| | International (Check here if [site] is not in the United States) | |
| 6d.1.3. | * Briefly describe the activities that will occur at [site]: The NBER is a funder through the NBER Roybal Center for Behavior Change in Health. No research will be performed to but they are requesting an IRB agreement. | there |
| 6d.1.4. | Determining Engagement: | |
| | Will [site] personnel conduct any of the following activities? | |
| | * 6d.1.4.1. Recruitment and Consent: | |
| | Inform potential participants of the availability of the research, provide study contact information, o seek permission for investigators to contact the potential participants? Yes No | r |
| | Obtain informed consent from the research participants? Yes No | |

\* 6d.1.4.2. Participant Data and Information:

Release to the study investigators data or information about the research participants that have been collected for non-research purposes?

Yes No

Obtain identifiable data or information about the research participants solely for the purposes of the research project?

https://istar.usc.edu/istar/sd/Doc/0/JGAV6OL8DC8UMQC1TH8OULIG00/fromString.html


AM

| UP-21-00030 | - COVID-19 ar | nd Preventive Health Behaviors | 4/29/21, 8:48 AN |
|---|---|---|---|
| | | Yes No | |
| | * 6d.1.4.3. | Participant Contact and Intervention: | |
| | | Interact with the research participants for routine care, follow up or commercial services? Yes No | |
| | | Interact or intervene with research participants for research purposes (including performing p or manipulating the environment)? Yes No | rocedures |
| * 6d.1.5 | | receive any direct federal support for this research? No | |
| Your an | swers indica | ate that [site] is engaged in the research. You must answer the following: | |
| 6d.1.6. | Does [site] Yes ( | have an IRB? No | |
| | 6d.1.6.1. | Will [site]'s IRB review this research? Yes No | |
| | * 6d.1.6.2. | Attach the IRB approval or, if [site] has elected to have USC/CHLA be the IRB of record, attach t authorization agreement. IAA - Jacobson Vaccination NBER Fully Executed.pdf(0.02) | he IRB |
| 6d.1.7. | Please pro | vide the following assurance: | |
| | | expected problems, protocol modifications, and interim results will be communicated to [site] an agencies (as applicable). | d |
| 6d.1.8. | Under which | IRB Authorization Agreement will [site] rely on the USC/CHLA IRB to review this study? | |
| | Other | | |
| 6d.1.9. | | the personnel at [site] carry out research activities such as obtaining consent or conducting stuss? (Deprecated Field - used to be 6c.1.3 only used for old studies) Yes No | dy |
| 6d.1.10. | [site] below | cate under which category(ies) [site] is engaged (see guidance) and attach a copy of the IRB appr<br>w. (Deprecated Field - old 6c.1.4 only used for old studies)<br>t Description | oval from |
| | | stitutions that receive an award through a grant, contract, or cooperative agreement directly from HHS for<br>pt human subjects research. | or the non- |
| | | stitutions whose employees or agents intervene for research purposes with any human subjects of the r<br>rming invasive or noninvasive procedures. | esearch by |
| | | stitutions whose employees or agents intervene for research purposes with any human subject of the rebulating the environment. | search by |

| UP-21-00030 - | - COVID-19 and Preventive Health Behaviors | 4/29/21, 8:48 AM |
|---|---|---|
| | (4) Institutions whose employees or agents interact for research purposes with any human subject of the re | search. |
| | (5) Institutions whose employees or agents obtain the informed consent of human subjects for the research | Ġ. |
| | (6) Institutions whose employees or agents obtain for research purposes identifiable private information or in biological specimens from any source for the research. | dentifiable |
| https://istar.use | c.edu/istar/sd/Doc/0/JGAV60L8DC8UMQC1TH8OULIG00/fromString.html | |

# Amended Protocol – April 2021 (0.05)

- Participants: Adult patients impaneled at Contra Costa Regional Medical Center (CCRMC) who are eligible for COVID-19 vaccination based on county and CCRMC determination.
  - Adults ages 18+, eligible for vaccination (as determined by the county)
  - Self-identified as African American/Black, White or Latino (irrespective of race).
  - Children are not included as they do not make their own health care decisions. We are interested in how adults make decisions about their own COVID-19 vaccination and other preventive health behaviors.
  - We are not explicitly studying a protected population. Prisoners are not impaneled at CCRMC. Pregnant women, to the extent they are not excluded in the county's vaccination plans, may be enrolled in the study. However, we will not explicitly target pregnant women or ask about pregnancy. Vaccination offers will be determined by medical personnel from the county and CCRMC, separate from the study.
- Recruitment Process (sampling strategy)
  - Eligible adults will be invited to participate in the study via email, mail, and/or text.
  - CCRMC will provide us with a list of impaneled adult patients who are eligible for vaccination based on county prioritization categories and individual health status and who self-identify as African American/Black, White or Latino (irrespective of race). The list will be shared by CCHS via USC Marshall's box.com accounts and will be managed by Tom Chang.
  - We will randomly sample and invite adults from this list to participate in a baseline survey. Recruitment in this way will continue until we reach a goal of 10,000 baseline survey responses.

# Enrollment Process

- Consent will occur through the baseline survey available via USC RedCAP and through the included consent documents.
- We will also ask for HIPAA authorization so that we can link the survey data to information on vaccinations.

# Methods

Our work will begin with a large online survey (N=10,000) of a random sample of the members of the county Medicaid managed care plan in Contra Costa County, CA. Contra Costa Health Plan (CCHP), has over 100,000 adult members. Over a quarter of adult members are Latino, a quarter non-Hispanic White and about 15% each are Black, Asian or of other/unknown race. Our sample will be drawn from CCHP members ages 18 and over who have not been previously vaccinated against COVID-19 and who have no contraindications to vaccination, as determined by county health plan medical staff. Because we are interested in testing race concordant messaging, we will also restrict to

members who are African American/Black, White or Latino (irrespective of race). Those of other/unknown race are excluded because they cannot be matched based on race to a messenger as are Asians because the group is comprised of populations that are both linguistically and culturally quite distinct. In particular, about a third of the "Asian" group is Filipino, a third Vietnamese, 25% Mandarin-speaking Chinese, 20% Cantonese-speaking Chinese, 15% Punjabi-speaking Indian, 10% Laotian, 10% Korean, and so on. As such, we do not think these populations can credibly be treated as one group for the purposes of studying race concordance and yet each group is individually too small to consider alone. Survey respondents will receive a \$5 gift card for their time and be entered into a raffle for a \$250 gift card.

In the survey, much of which we have previously piloted for a related project, we will capture rates of preventive health behaviors, including mask-wearing, hand washing, and, most importantly, willingness to vaccinate. Stratifying based on race/ethnicity, age-group and other characteristics predictive of vaccine take-up, we will randomize the 10,000 respondents to one of four arms:

- 1. Control arm [2,500]
- 2. Messaging/Information Arm 1: no information/emotional message [N=2,500]
- 3. Messaging/Information Arm 2: safety and effectiveness information [N=2,500]
- 4. Messaging/Information Arm 3: information on consequences of going unvaccinated].

Figure. Randomization Design



The information arms have been designed with the experimental literature on vaccination intentions in mind (see Brewer et al. 2017 for a review). That literature finds, among other things, that

messages aimed at clarifying the negative outcomes of not getting vaccinated are much more effective at changing intentions than messages that try to correct misperceptions about vaccine safety. Within the arm 3 and arm 4 message groups, we will further randomize participants to race/ethnicity concordant/discordant video messages and to gender concordant/discordant messages. This intervention builds on recent evidence that race-concordant health care providers increase health screening take-up (Alsan et al. 2019).

Each of these four arms will be interacted with a financial incentive of \$10 (N=2,500) or \$50 (N=2,500) and, separately with a convenient link to the county public vaccine appointment scheduling system highlighted for participants (N=5,000).

The above treatments are designed to test the role of the following on vaccine take-up:

- Financial incentives [N=5,000] vs. no financial incentives [N=5,000]
  - 2,500 will be randomized to a \$10 incentive and 2,500 to a \$50 incentive

- Convenient scheduling link highlighted [N=5,000] vs. not [N=5,000]
- Messaging [N=7,500] vs not [2,500]
  - Message type: emotion [N=2,500] vs. safety and effectiveness [N=2,500]
     vs. consequences of not vaccinating [N=2,500]
- Race concordant [N=2,500] vs. race discordant messenger [N=2,500]
- Gender concordant [N=2,500] vs. gender discordant messenger [N=2,500]

These financial incentives of \$10 or \$50 are in line with the prior literature. For example, Bronchetti, Huffman, and Magenheim (2015) paid college students \$30 for flu vaccinations in 2012. In addition, the \$50 incentive is in-line with 2 hours of time at the minimum wage plus transportation costs. These incentives will be paid for with funding from J-PAL. While financial incentives for vaccination have faced some criticism (Largent and Miller 2021), prior work suggests small incentives can be quite effective (Bronchetti, Huffman, and Magenheim 2015). Given the urgency of the issue, we think it is crucial to test the effectiveness of financial incentives against other potential tools to improve vaccine take-up. We will also examine study impacts for subpopulations of interest identified in our baseline survey (e.g., groups at a high risk for adverse health outcomes or young adults who have high potential to be super-spreaders of COVID-19).

We understand that the IRB is concerned that the incentives for vaccination are not equal across participants in the incentive arm. However, this approach is fairly standard in behavioral economic studies and has been approved by many IRBs at peer institutions. We highlight just a few such health studies here but there are dozens of other relevant examples:

- Alsan et al. (2019), which studied preventive health care among African American men, included a condition that randomly offered subjects incentives of \$5 or \$10 for selecting an influenza vaccination. These rewards were for intentions and were irrespective of actual vaccination. This study was approved by Stanford's IRB. The protocol is available in Alsan et al. (2018) https://doi.org/10.1257/rct.2497-2.0.
- 2. Bachireddy et al. (2019), which studied physical activity, compared 3 different 2-week incentive programs with rewards for daily steps taken. Incentives varied from \$0.10 per 10,000 steps to \$2 per 10,000 steps, a 20-fold difference, over the 2-week intervention period. This study was approved by the IRB at University of Pennsylvania.
- 3. Jones et al. (2019), which studied workplace wellness programs, offered varying levels of cash rewards (\$100 vs. \$200) to University of Illinois employees for completing a biometric screening and health risk assessment and an additional cash reward for completing each wellness activity (\$25 vs. \$75). The study was approved by the IRBs at University of Illinois Urbana Champaign, the University of Chicago and the National Bureau of Economic Research.

We believe our work is in line with these and many other studies. It is also extremely policy relevant given concern about vaccine take-up.

Our primary outcomes are vaccine take-up at one month and vaccine intentions at the time of survey. Secondary analysis will consider any vaccine take-up over longer time periods.

Overview of procedures to be used for

- Data collection tools
  - Baseline survey Survey will be translated into Spanish and thus available in both Spanish and English for respondents to choose from in RedCAP.
  - Administrative data from CCRMC on COVID-19 tests, vaccinations, hospitalizations
- Vaccination appointments in Contra Costa have been open to all age groups since March 30, 2021.
- Research procedures will end once survey respondents have "received" an intervention. The research team will not take part in any delivery of care. Thus, any actual take-up of vaccinations will be subject to normal CCHS standard of care.
- Data Analysis

# Randomization

Randomization will be performed in the RedCAP system. In practice, the randomization will divide the sample into 60 possible conditions:

- 1. Control [N=625]
- 2. Control x \$10 financial [N=312.5]
- 3. Control x \$50 financial [N=312.5]
- 4. Control x link [N=625]
- 5. Control x \$10 financial x link [N=312.5]
- 6. Control x \$50 financial x link [N=312.5]
- 7. No information/Emotional (language concordant) [N=625]
- 8. No information/Emotional (language concordant) x \$10 financial [N=312.5]
- 9. No information/Emotional (language concordant) x \$50 financial [N=312.5]
- 10. No information/Emotional (language concordant) x link [N=625]
- 11. No information/Emotional (language concordant) x \$10 financial x link [N=312.5]
- 12. No information/Emotional (language concordant) x \$50 financial x link [N=312.5]
- 13. Safety and effectiveness (race concordant, male) [N=156.25]
- 14. Safety and effectiveness (race concordant, male) x \$10 financial incentive [N=78.125]
- 15. Safety and effectiveness (race concordant, male) x \$50 financial incentive [N=78.125]
- 16. Safety and effectiveness (race concordant, male) x link [N=156.25]

- 17. Safety and effectiveness (race concordant, male) x \$10 financial incentive [N=78.125]
- 18. Safety and effectiveness (race concordant, male) x \$50 financial incentive [N=78.125]
- 19. Safety and effectiveness (race concordant, female) [N=156.25]
- 20. Safety and effectiveness (race concordant, female) x \$10 financial incentive [N=78.125]
- 21. Safety and effectiveness (race concordant, female) x \$50 financial incentive [N=78.125]
- 22. Safety and effectiveness (race concordant, female) x link [N=156.25]
- 23. Safety and effectiveness (race concordant, female) x \$10 financial incentive x link [N=78.125]
- 24. Safety and effectiveness (race concordant, female) x \$50 financial incentive x link [N=78.125]
- 25. Safety and effectiveness (race discordant, male) [N=156.25]
- 26. Safety and effectiveness (race discordant, male) x \$10 financial incentive [N=78.125]
- 27. Safety and effectiveness (race discordant, male) x \$50 financial incentive [N=78.125]
- 28. Safety and effectiveness (race discordant, male) x link [N=156.25]
- 29. Safety and effectiveness (race discordant, male) x financial incentive x link [N=78.125]
- 30. Safety and effectiveness (race discordant, male) x financial incentive x link [N=78.125]
- 31. Safety and effectiveness (race discordant, female) [N=156.25]
- 32. Safety and effectiveness (race discordant, female) x \$10 financial incentive [N=78.125]
- 33. Safety and effectiveness (race discordant, female) x \$50 financial incentive [N=78.125]
- 34. Safety and effectiveness (race discordant, female) x link [N=156.25]
- 35. Safety and effectiveness (race discordant, female) x \$10 financial incentive x link [N=78.125]
- 36. Safety and effectiveness (race discordant, female) x \$50 financial incentive x link [N=78.125]
- 37. Consequences of going unvaccinated (race concordant, male) [N=156.25]
- 38. Consequences of going unvaccinated (race concordant, male) x \$10 financial incentive [N=78.125]
- 39. Consequences of going unvaccinated (race concordant, male) x \$50 financial incentive [N=78.125]
- 40. Consequences of going unvaccinated (race concordant, male) x link [N=156.25]
- 41. Consequences of going unvaccinated (race concordant, male) x \$10 financial incentive x link [N=78.125]

- 42. Consequences of going unvaccinated (race concordant, male) x \$50 financial incentive x link [N=78.125]
- 43. Consequences of going unvaccinated (race concordant, female) [N=156.25]
- 44. Consequences of going unvaccinated (race concordant, female) x \$10 financial incentive [N=78.125]
- 45. Consequences of going unvaccinated (race concordant, female) x \$50 financial incentive [N=78.125]
- 46. Consequences of going unvaccinated (race concordant, female) x link [N=156.25]
- 47. Consequences of going unvaccinated (race concordant, female) x \$10 financial incentive x link [N=78.125]
- 48. Consequences of going unvaccinated (race concordant, female) x \$50 financial incentive x link [N=78.125]
- 49. Consequences of going unvaccinated (race discordant, male) [N=156.25]
- 50. Consequences of going unvaccinated (race discordant, male) x \$10 financial incentive [N=78.125]
- 51. Consequences of going unvaccinated (race discordant, male) x \$50 financial incentive [N=78.125]
- 52. Consequences of going unvaccinated (race discordant, male) x link [N=156.25]
- 53. Consequences of going unvaccinated (race discordant, male) x \$10 financial incentive x link [N=78.125]
- 54. Consequences of going unvaccinated (race discordant, male) x \$50 financial incentive x link [N=78.125]
- 55. Consequences of going unvaccinated (race discordant, female) [N=156.25]
- 56. Consequences of going unvaccinated (race discordant, female) x \$10 financial incentive [N=78.125]
- 57. Consequences of going unvaccinated (race discordant, female) x \$50 financial incentive [N=78.125]
- 58. Consequences of going unvaccinated (race discordant, male) x link [N=156.25]
- 59. Consequences of going unvaccinated (race discordant, male) x \$10 financial incentive x link [N=78.125]
- 60. Consequences of going unvaccinated (race discordant, male) x \$50 financial incentive x link [N=78.125]

# Protection of Data

All identifiable data (names and either phone, email or physical address) will be available only for the purposes of 1) inviting study participants and 2) linking data. These data will be kept on secure password-protected USC Marshall servers and will only be accessible to Drs. Chang and Pramanik. Data sharing will occur through Marshall administered Box accounts. Box encrypts data at rest and in transit. Tom Chang will handle all matching of surveys and administrative data.

Name and address information, not linked to any health information, will also be made available to the minimum number of research staff needed to invite participants to our surveys.

Analytic datasets available to the research team will be limited datasets, without name, address, or any contact information. That data will be stored in a password protected shared study drive.

# References

Alsan, Marcella, Owen Garrick and Grant Graziani. 2018. "The Oakland Men's Health Disparities Study." AEA RCT Registry. March 21. https://doi.org/10.1257/rct.2497-2.0

Alsan M., Owen G. and Graziani G. 2019. "Does Diversity Matter for Health? Experimental Evidence from Oakland." *American Economic Review* 109(12): 4071-4111. DOI: 10.1257/aer.20181446.

Bachireddy C, Joung A, John LK, et al. 2019. Effect of Different Financial Incentive Structures on Promoting Physical Activity Among Adults: A Randomized Clinical Trial. *JAMA Netw Open.* 2019;2(8):e199863. doi:10.1001/jamanetworkopen.2019.9863

Bronchetti ET, Huffman DB and Magenheim E. 2015. Attention, intentions, and follow-through in preventive health behavior: Field experimental evidence on flu vaccination. Journal of Economic Behavior & Organization, 116, 270–291. DOI: 10.1016/j.jebo.2015.04.003.

Damon Jones, David Molitor, Julian Reif, 2019. What do Workplace Wellness Programs do? Evidence from the Illinois Workplace Wellness Study, The Quarterly Journal of Economics, 134(4): 1747-1791 qjz023, https://doi.org/10.1093/qje/qjz023

Largent EA, FG Miller. 2021. Problems With Paying People to Be Vaccinated Against COVID-19

JAMA Published online January 6, 2021. PMID: 33404585

UP-21-00030-AM002 - Increase survey incentive

6/1/21, 5:13 PM

Version: 1.1

Application Version Date: 6/1/2021

Date: Tuesday, June 1, 2021 4:21:06 PM Print Close

# 1. Project Identification Information

| 1. I Toject Identification information | | |
|---|---|---|
| Title of the Protocol: COVID-19 and Preventive Health Behaviors (UP-21-00030) | | |
| Principal Investigator: Mireille Jacobson | | |
| Study Coordinator: | | |
| AM1.1. | * Identifier for this Amendment: Increase survey incentive | |
| AM1.2. | * Type of Amendment(s) (check a | ill that apply): |
| | Туре | 2 00 0000 |
| | ☐ Editorial | |
| | Drug or Device | |
| | Enrollment Status Change | |
| | Funding | |
| | ☐ Informed Consent and/or Add | lenda |
| | ☐ Investigator's Brochure / Pack | kage Insert |
| | Locations | |
| | Number of Subjects | |
| | Procedures and/or Protocol | |
| | Recruitment Materials | |
| | Risks/Harms | |
| | Study Personnel | |
| | Subject Population | |
| | Subject Reimbursement / C | ompensation |

https://istar.usc.edu/istar/sd/Doc/0/0J254JE3608UMQK1TH80ULIG00/fromString.html

Page 1 of 2

| 1-00030 | 00-AM002 - Increase survey incentive | 6 <i> </i> 1/21, |
|---|---|---|
| | ☐ Other | |
| AM1.: | 3. Will the changes you are making affect the accuracy of the study abstract? Yes No | |
| AM1.6 | 6. Has the risk/benefit ratio changed? Yes No | |
| 14. | Subject Reimbursement / Compensation | |
| | screen is required if you indicated this amendment involves changes to Subject Reimbursement or pensation policies or amounts. (Question 1.2.) | |
| \<br>( | Please describe each of the changes to Subject Reimbursement and/or Compensation and provide a rationale for the change. We would like to increase our survey incentive to \$25 to address low take-up. We have included consent documents in both English and Spanish for a \$25 survey incentive. We have made no changes to the study design itself. | |
| Modif<br>effect | must make your changes in the body of the main study application by clicking on "Edit ified Study" in the Amendment workspace. Please remember to revise any other information sted by this change. It is likely that changes to subject compensation will require updating sent documents (item 24). | |
| 99. | Modified Study Link | 18 |
| | ake your changes to the study specified in this amendment, please: | |
| To ma | | _ |
| To ma | ake your changes to the study specified in this amendment, please: | |
| To ma<br>1.<br>2.<br>3. | ake your changes to the study specified in this amendment, please: Click the Finish button in the menu bar above or below this form. | |

# **APPENDIX B: Informed Consent Documents and HIPAA Authorization**

University of Southern California USC Davis School of Gerontology 3715 McClintock Ave, Los Angeles, CA 90089

## INFORMED CONSENT FOR RESEARCH

Study Title: COVID-19 and Preventive Health Behaviors

Principal Investigator: Mireille Jacobson, Ph.D.

Department: USC Leonard Davis School of Gerontology

# INTRODUCTION

We invite you to take part in a research study. Please take as much time as you need to read the consent form. You may want to discuss it with your family, friends, or your personal doctor. If you find any of the language difficult to understand, please ask questions. You can contact the study lead, Mireille Jacobson by phone or email: tel: 213-986-6076 or email: mireillj@usc.edu. If you decide to participate, you will be asked to sign this form. A copy of the signed form will be provided to you for your records.

# **KEY INFORMATION**

The following is a short summary of this study to help you decide whether you should participate. More detailed information is listed later in this form.

- 1. Being in this research study is voluntary-it is your choice.
- You are being asked to take part in this study so that Contra Costa County can
  better understand COVID-19 vaccine uptake. The purpose of this study is to
  analyze behaviors in relation to COVID-19, including vaccinations. Procedures will
  include the completion of a baseline survey. Your participation in the baseline
  survey will last approximately 15 minutes and is completely voluntary.
- 3. If you consent to be part of this study, information on health care, received at Contra Costa Regional Medical Center (CCRMC) or otherwise provided by Contra Costa Health Services or the County of Contra Costa, including COVID-19 tests and test results and COVID-19 vaccination status, may be shared with the study investigators. The investigators will keep your data secure and will not share your information with anyone outside the study team. All your information will be kept confidential.
- 4. Some people who participate in this study will be randomly selected to receive additional information about COVID-19 vaccines. Some people who participate will be randomly selected to receive gift certificates for being vaccinated that vary between \$10 and \$50. We will contact you if you are selected for either of these.
- 5. There are risks from participating in this study. The most common risks are that some of the survey questions may make the participant feel uneasy or embarrassed. There is also a small risk that people not connected with the study will learn the participants identity or their personal information. More detailed

Version Date: May 26, 2021 

information about the risks of this study can be found under the "Risk and Discomfort" section.

- 5. You may not receive any direct benefit from taking part in this study. However, your participation in this study may help us learn how to better manage the COVID-19 pandemic in Contra Costa County.
- 6. If you decide not to participate in this research, your other choices may include: not participate in the study.

# **DETAILED INFORMATION**

# **PURPOSE**

The purpose of this study is to better understand COVID-19 vaccinations and other preventive behaviors taken to mitigate the spread of the disease. This research is designed to help Contra Costa better understand the COVID-19 pandemic and shape and improve its efforts to better serve the community. About 10,000 participants will take part in the study.

# **PROCEDURES**

If you decide to take part, you will be asked to complete a baseline survey on your phone, tablet or internet connected computer. The surveys take about 15 minutes to complete. The surveys ask you about COVID-19, how it has affected your day to day life, as well as about your life more generally. Your survey responses may be linked to your COVID-19 test and vaccination information and possibly other data already captured by the county health system. However, all your information will remain confidential and will be anonymized for research purposes.

- 1. You will complete a 15-minute baseline survey.
- 2. Your survey data may be linked to data from Contra Costa Health Services and shared with the study investigators.
- 3. Some people who participate will be randomly selected to receive additional information about the COVID-19 vaccine.
- 4. Some people who participate will be randomly selected to receive gift certificates for being vaccinated of \$10 or \$50. We will contact you if you are selected for these.

# **RISKS AND DISCOMFORTS**

Possible risks and discomforts you could experience during this study include:

**Surveys/Questionnaires/Interviews:** Some of the questions may make you feel uneasy or embarrassed. You can choose to skip or stop answering any questions you don't want to.


**Breach of Confidentiality:** There is a small risk that people who are not connected with this study will learn your identity or your personal information.

# **BENEFITS**

There are no direct benefits to you from taking part in this study. However, your participation in this study may help us learn more about the current COVID-19 (coronavirus) pandemic in Contra Costa County to improve county-wide efforts to contain the virus.

# PRIVACY/CONFIDENTIALITY

We will keep your records for this study confidential as far as permitted by law. However, if we are required to do so by law, we will disclose confidential information about you. Efforts will be made to limit the use and disclosure of your personal information, including research study and medical records, to people who are required to review this information. Information about this study will be posted at ClinicalTrials.gov. We may publish the information from this study in journals or present it at meetings. We will not use your name on ClinicalTrials.gov, in any journal articles, or in any meeting presentations.

The University of Southern California's Institutional Review Board (IRB) may review your records. Organizations that may also inspect and copy your information include: the Contra Costa County Regional Medical Center's Institutional Review Committee (IRC) and the National Bureau of Economic Research's IRB. The IRB/IRC reviews and monitors research studies to protect the rights and welfare of research subjects.

Your information that is collected as part of this research will be used or distributed for future research studies without your additional informed consent. Any information that identifies you (such as your name) will be removed from your private information before being shared with others.

## **ALTERNATIVES**

An alternative would be to not participate in this study.

# **PAYMENTS**

If you complete the baseline survey, you will receive a gift card of \$25 for your time and be entered into a drawing for a \$250 gift card. In total, we will raffle off 20 gift cards valued at \$250 each. Some people who participate will be randomly selected to receive gift certificates for being vaccinated between \$10 and \$50.

# COST


# Study ID: UP-21-00030 Valid From: 6/1/202

# University of Southern California USC Davis School of Gerontology 3715 McClintock Ave Los Angeles, CA 90089

There are no costs related to participation.

# **VOLUNTARY PARTICIPATION**

It is your choice whether to participate. If you choose to participate, you may change your mind and leave the study at any time. Refusal to participate or stopping your participation will involve no penalty or loss of benefits to which you are otherwise entitled.

If you stop being in the research, already collected data may not be removed from the study database. You will be asked whether the investigator can continue to collect data from your records. If you agree, this data will be handled the same as the research data. No new information will be collected about you or from you by the study team without your permission.

Your personal information, including any identifiable information, that has already been collected up to the time of your withdrawal will be kept and used to guarantee the integrity of the study, to determine the safety effects, and to satisfy any legal or regulatory requirements.

# **CONTACT INFORMATION**

If you have questions, concerns, complaints, or think the research has hurt you, talk to the study investigator at

Mireille Jacobson, tel: 213-986-6076 or email: mireillj@usc.edu

This research has been reviewed by the USC Institutional Review Board (IRB). The IRB is a research review board that reviews and monitors research studies to protect the rights and welfare of research participants. Contact the IRB if you have questions about your rights as a research participant or you have complaints about the research. You may contact the IRB at (323) 442-0114 or by email at irb@usc.edu.

# STATEMENT OF CONSENT

| I have read (or someone has read to me) the information provided above. I have been |
|---|
| given a chance to ask questions. All my questions have been answered. By signing this |
| form, I am agreeing to take part in this study. |

| 0.607 | • | • | • | - |
|----------|---------|-----------|-----------|---|
| □ I agre | e to pa | rticipate | | |
| □IdoN | IOT agr | ee to pa | rticipate | |


Study Title: COVID-19 and Preventive Health Behaviors

IRB#: UP-21-00030

# HIPAA AUTHORIZATION TO USE CONTRA COSTA HEALTH SERVICES (CCHS) HEALTH INFORMATION FOR RESEARCH

# 1. Purpose of this Form:

A federal law known as the Health Insurance Portability and Accountability Act (HIPAA) protects how your health information is used. HIPAA generally does not allow your health information to be used or released for research purposes without your written permission. Health information protected under the law includes: medical and dental records, bills or other payment records for health care received, tissue samples, x-rays, laboratory results and any other health information that identifies you. State laws also protect how your health information may be used.

By signing this form, you are allowing your health care providers (for example, physicians, dentists, hospitals, clinics) to share your health information with the researchers and others involved in this research study for the uses described below and also described in the informed consent.

# 2. Who May Release Your Health Information:

This document permits (i) Contra Costa Health Services to release health information about you to (ii) the researchers for the research purposes described in this document and the informed consent.

# 3. What Health Information Will Be Used:

Contra Costa Health Services is permitted to use and release (i) all health information that is created during this research study; and all of your health information that the health care provider has in his or her possession, but does <u>not</u> include HIV test results, mental health diagnosis and treatment records, and drug or alcohol treatment records.

# 4. How Your Health Information Will Be Used:

Your health information may be shared with the following individuals or entities for the following purposes:

Study Title: COVID-19 and Preventive Health Behaviors

IRB #: UP-21-00030

Researchers (those individuals in charge of the study), research staff, and students to conduct the research described in the informed consent and other activities related to the research, such as conducting safety analyses.

- The research sponsors, J-PAL North America and the National Bureau of Economic Research, and their authorized representatives, business partners, clinical research organizations and affiliates for the purposes described in the informed consent and for other activities related to the research, such as assessing the safety or efficacy of the drug, device or treatment included in the study, improving designs of future studies or obtaining approval for new drugs, devices or health care products.
- The USC Institutional Review Boards that review research involving human subjects in accordance with regulations;
- USC's clinical trial organization that supports clinical trials administration at USC,
- Other USC offices involved in regulatory compliance, including the Offices of General Counsel and Compliance,
- U.S. government agencies, such as the Food and Drug Administration and the Office for Human Research Protections, government agencies from other countries, and others who are authorized by law to review or oversee this research.

# 5. Creation of a Research Database:

The following is an optional research activity. You can choose whether or not to participate in these activities and it will not affect your ability to participate in the main research study. Please initial on the line below to give your specific permission to this activity.

Researchers will often study existing health information from large groups of patients in order to test or validate theories that the researcher develops. By initialing above, you allow the USC research team to put your health information in a research database or repository for future research purposes. The USC Institutional Review Board still may review how the researcher uses or releases your health information for future research purposes.

2

Study Title: COVID-19 and Preventive Health Behaviors

IRB#: UP-21-00030

This section of the Authorization will remain in effect indefinitely unless you revoke (cancel) it as described below.

# 6. Scope of this Authorization:

The USC research team will use and release your health information for the purposes described in this authorization and the informed consent or as otherwise permitted by law. However, health information that is shared with others outside USC may not be protected by HIPAA once it is released. Certain health information may still be protected under state law.

# 7. Right to Deny Access to Health Information:

You may not be permitted to access (review or copy) your health information created during this research study while the research study is in progress. You may be entitled to access your health information once the research study is completed.

# 8. Term of this Authorization:

Except for database research, this authorization expires 25 years from the date the study is completed or terminated.

# 9. Refusal to Sign/Right to Revoke:

You must sign this Authorization in order to participate in this research. You may change your mind and revoke (withdraw or cancel) this authorization and your participation in this research study at any time. To do so, your revocation must be sent in writing to the Principal Investigator and include: (1) the title of the research study; and (2) your name and telephone number or address. Please send the revocation to the following:

Professor Mireille Jacobson 3715 McClintock Ave

Los Angeles, CA 90089

You will not be permitted to participate in the research and health information that identifies you will no longer be collected as of the date the Principal Investigator receives

Study Title: COVID-19 and Preventive Health Behaviors

IRB#: UP-21-00030

your revocation. However, we may still use and share health information about you that has already been obtained as necessary in order to maintain the integrity of the research study. Also, if the law requires it, the researchers, sponsor, and government agencies may continue to look at your records to review the quality or safety of the study.

4

Study Title: COVID-19 and Preventive Health Behaviors

IRB#: UP-21-00030

# 10. Questions Regarding Your Privacy Rights:

Please contact the USC Office of Compliance by telephone at 213-740-8258 or email at <a href="mailto:compliance@usc.edu">compliance@usc.edu</a> if you have questions about your privacy rights.

# Agreement:

I have read (or someone has read to me) the information provided above. I have been given the opportunity to ask questions and all of my questions have been answered to my satisfaction. By signing below, I agree that my health information may be used as described in this form.

| Name of Participant | Signature | Date Signed |
|---------------------|-----------|-------------|

Rev 10.16 5

# AUTORIZACIÓN PARA PARTICIPAR EN UN ESTUDIO DE INVESTIGACIÓN

Título del estudio: COVID-19 y Comportamiento de Salud Preventivos

Investigadora principal: Mireille Jacobson, Ph.D.

**Departamento: USC Leonard Davis School of Gerontology** 

## INTRODUCCIÓN

Te invitamos a participar en un estudio de investigación. Tómate el tiempo que necesites para leer el formulario de consentimiento. Es posible que desees discutirlo con tu familia, amigos o tu médico personal. Si encuentras que alguno de los idiomas es difícil de entender y tienes dudas, puedes comunicarte con la directora del estudio, Mireille Jacobson, por teléfono o correo electrónico: 213-986-6076 o correo electrónico: mireillj@usc.edu. Si decides participar, se te pedirá que firmes este formulario. Se te proporcionará una copia del formulario firmado para tus registros.

# INFORMACIÓN IMPORTANTE

El siguiente es un breve resumen de este estudio para ayudarte a decidir si quieres participar. Información detallada encontraras más adelante en este formulario.

- 1. Es totalmente voluntario participar en este estudio, simplemente es tu elección.
- 2. Se te está pidiendo que participes en este estudio para que el Condado de Contra Costa pueda entender mejor el comportamiento de la vacunación COVID-19. El propósito de este estudio es analizar los comportamientos en relación con COVID-19, incluidas las vacunas. Los procedimientos incluirán la realización de una encuesta. Tú participación en este estudio durará aproximadamente 15 minutos y es totalmente voluntario.
- 3. Si aceptas formar parte de este estudio, la información sobre la atención médica, recibida en el Centro Médico Regional de Contra Costa (CCRMC) o proporcionada de otra manera por Contra Costa Health Services o el Condado de Contra Costa incluidas las pruebas COVID-19 y los resultados de las pruebas y COVID -19 estado de vacunación, se puede compartir con los investigadores del estudio. Los investigadores mantendrán tus datos seguros y no compartirán tu información con nadie fuera del equipo del estudio. Toda tu información se mantendrá confidencial.
- 4. Algunas personas que participan en este estudio serán seleccionadas al azar para recibir información adicional sobre las vacunas COVID-19. Algunas personas que participen serán seleccionadas al azar para recibir una tarjeta de regalo por ser vacunados que varían entre \$10 y \$50. Nos comunicaremos contigo si eres seleccionado para alguno de estos.


- 5. Existen algunos riesgos por participar en este estudio. Los riesgos más comunes son que algunas preguntas de la encuesta pueden hacer que el participante se sienta incómodo o avergonzado, y existe un pequeño riesgo de que algunas personas que no están relacionadas con el estudio conozcan la identidad de los participantes o su información personal.
- 5. Tú participación en este estudio puede ayudarnos a aprender cómo manejar mejor la pandemia de COVID-19 en el Condado de Contra Costa.
- 6. Si decides no participar en esta investigación, puedes simplemente no participar en el estudio.

# INFORMACIÓN DETALLADA

# **PROPÓSITO**

El propósito de este estudio es comprender mejor las vacunas COVID-19 y los comportamientos adoptados para mitigar la propagación de la enfermedad. Está investigación está diseñada para ayudar a Contra Costa a comprender mejor la pandemia de COVID-19 y dar forma y mejorar sus esfuerzos para servir mejor a la comunidad. Alrededor de 10.000 participantes participarán en el estudio.

# **PROCEDIMIENTOS**

Si decides participar, se te pedirá que completes una encuesta en tú teléfono, tableta o computadora conectada a Internet. Las encuestas tardan entre 15 minutos en completarse. Las encuestas te preguntan sobre COVID-19, cómo te ha afectado tu vida cotidiana, así como sobre tu vida en general. Las respuestas de tu encuesta pueden estar vinculadas a la información de tu pruebas de COVID-19 y la información de vacunacíon y posiblemente a otros datos ya capturados por el sistema de salud del condado. Sin embargo, toda tu información permanecerá confidencial y se mantendrá anónima para fines de investigación.

- 1. Completarás una encuesta inicial de 15 minutos.
- 2. Los datos de tu encuesta pueden estar vinculados a datos de Contra Costa Health Services y compartidos con los investigadores del estudio.
- 3. Algunas personas que participen en este estudio serán seleccionadas al azar para recibir información adicional sobre las vacunas COVID-19.
- 4. Algunas personas que participen serán seleccionadas al azar para recibir una tarjeta de regalo por ser vacunados que varían entre \$10 y \$50. Nos comunicaremos contigo si eres seleccionado para alguno de estos.

# **RIESGOS E INCOMODIDADES**


Los posibles riesgos y molestias que podrías experimentar durante este estudio incluyen:

**Encuestas/ Cuestionarios/ Entrevistas:** algunas de las preguntas pueden hacerte sentir incómodo o avergonzado. Puedes optar por omitir o dejar de responder cualquier pregunta que no desees.

**Incumplimiento de la confidencialidad**: existe un pequeño riesgo de que algunas personas que no están relacionadas con este estudio conozcan tu identidad o tu información personal.

## **BENEFICIOS**

No hay beneficios directos para ti al participar en este estudio. Sin embargo, tu participación en este estudio puede ayudarnos a aprender más sobre la pandemia actual de COVID-19 (coronavirus) en el Condado de Contra Costa para mejorar los esfuerzos de todo el condado para contener el virus.

# PRIVACIDAD / CONFIDENCIALIDAD

Mantendremos la confidencialidad de tus registros para este estudio hasta donde lo permita la ley. Sin embargo, si la ley nos exige hacerlo, divulgaremos información confidencial sobre tí. Se realizarán esfuerzos para limitar el uso y la divulgación de tu información personal, incluidos el estudio de investigación y los registros médicos, a las personas que deben revisar esta información. La información sobre este estudio se publicará en ClinicalTrials.gov. Podemos publicar la información de este estudio en revistas o presentarla en reuniones. No usaremos tu nombre en ClinicalTrials.gov, en ningún artículo de revista o en presentaciones de reuniones..

La Junta de Revisión Institucional (IRB) de la Universidad del Sur de California puede revisar tus registros. Las organizaciones que también pueden inspeccionar y copiar tu información incluyen: el Comité de Revisión Institucional (IRC) del Centro Médico Regional del Condado de Contra Costa y la IRB del National Bureau of Economic Research (NBER). El IRB / IRC revisa y supervisa los estudios de investigación para proteger los derechos y el bienestar de los sujetos de investigación.

Tu información que se recopilará como parte de esta investigación se utilizará o distribuirá para futuros estudios de investigación sin tu consentimiento adicional. Cualquier información que te identifique (como tu nombre) será eliminada de su información privada o muestras antes de ser compartida con otros.

# **ALTERNATIVAS**

Una alternativa sería no participar en este estudio.


# **Pagos**

Recibirá una tarjeta de regalo de \$25 por la encuesta y entrarás a una rifa de \$250 en una tarjeta de regalo. En total, sortearemos 20 tarjetas de regalo valoradas en \$250 cada una. Algunas personas que participen serán seleccionadas al azar para recibir una tarjeta de regalo por ser vacunados que varían entre \$10 y \$50.

# COSTO

No hay costos relacionados con la participación.

# PARTICIPACION VOLUNTARIA

Es tu elección participar. Si eliges participar, puedes cambiar de opinión y abandonar el estudio en cualquier momento. Negarse a participar o suspender tu participación no implicará penalización o pérdida de beneficios a los que tiene derecho de otra manera.

Si dejas de participar en la investigación, es posible que los datos ya recopilados no se eliminen de la base de datos del estudio. Se te preguntará si el investigador puede continuar recopilando datos de tus registros. Si estás de acuerdo, estos datos se manejarán igual que los datos de la investigación. El equipo del estudio no recopilará información o muestras nuevas sobre ti o de ti sin tu permiso.

Puede ser que el estudio, después de que hayas decidido dejarlo, necesite comunicarte de cualquier evento de seguridad que pueda haber experimentado debido a tu participación a todas las entidades involucradas en el estudio. Tu información personal, que incluya cualquier información que te pueda identificar, y que se haya recopilado hasta el momento de tu retiro, se conservará y utilizará a para garantizar la integridad del estudio, determinar los efectos de seguridad y satisfacer cualquier requisito legal o reglamentario.

# INFORMACIÓN DEL CONTACTO

Si tienes preguntas, inquietudes, quejas o crees que la investigación te ha perjudicado, habla con la investigadora del estudio:

Mireille Jacobson, tel: 213-986-6076 o correo electrónico: mireilli@usc.edu

Esta investigación ha sido revisada por la Junta de Revisión Institucional (IRB) de la USC. El IRB es una junta de revisión de investigación que revisa y monitorea los estudios de investigación para proteger los derechos y el bienestar de los participantes de la investigación. Ponte en contacto con el IRB si tienes preguntas sobre tus derechos como participante de la investigación o si tienes quejas sobre la investigación.


# Study ID: UP-21-00030 Valid From: 6/1/2021

# University of Southern California USC Davis School of Gerontology 3715 McClintock Ave., Los Angeles, CA 90089

Puede comunicarse con el IRB al (323) 442-0114 o por correo electrónico a irb@usc.edu.

# **DECLARACIÓN DE CONSENTIMIENTO**

He leído (o alguien me ha leído) la información proporcionada anteriormente. Se me ha dado la oportunidad de hacer preguntas. Todas mis preguntas han sido respondidas. Al firmar este formulario, acepto participar en este estudio.

| ☐ Acepto | participar |
|----------|------------|

☐ NO estoy de acuerdo en participar


Título del estudio: COVID-19 y Comportamiento de Salud Preventivos

N.° IRB. UP-21-00030

# AUTORIZACIÓN DE CONSENTIMIENTO CON LA LEY HIPAA PARA UTILIZAR INFORMACIÓN DE SALUD DE CONTRA COSTA HEALTH SERVICES CON FINES DE INVESTIGACIÓN

# 1. Finalidad de este formulario:

La ley federal denominada Ley de Portabilidad y Responsabilidad de Seguros de Salud (HIPAA, por sus siglas en inglés) protege la forma en que se utiliza su información de salud. Por lo general, la ley HIPAA no permite que su información de salud se utilice o divulgue con fines de investigación sin su autorización por escrito. La información sobre la salud protegida por la ley incluye: historias clínicas o registros dentales, facturas u otros registros de pago por atención de salud recibida, muestras de tejido, radiografías, resultados de análisis clínicos y cualquier otra información de salud que lo identifique como persona. Las leyes estatales también protegen el modo en que se puede utilizar su información de salud.

Mediante su firma en este formulario, usted autoriza a sus proveedores de atención de salud (por ejemplo, médicos, dentistas, hospitales, clínicas) a compartir su información de salud con los investigadores y demás personas que formen parte de este estudio de investigación para los usos que se detallan a continuación y que también se describen en el consentimiento informado.

# 2. Quién puede difundir su información de salud:

Este documento permite que (i) Contra Costa Health Services a continuación difundan información de salud sobre usted con (ii) los investigadores de los fines de investigación descritos en este documento y en el consentimiento informado:

Título del estudio: COVID-19 y Comportamiento de Salud Preventivos

N.° IRB. UP-21-00030

# 3. Qué información de salud se utilizará:

Contra Costa Health Services tienen permiso para utilizar y divulgar (i) toda la información de salud que se cree durante este estudio de investigación, y toda la información de salud que el proveedor de atención de salud tenga en su posesión, pero que no incluye resultados sobre la prueba del VIH, registros de diagnósticos y tratamientos de salud mental ni registros de tratamientos por alcohol o drogas

# 4. De qué manera se utilizará su información de salud:

Es posible que su información de salud se comparta con las siguientes personas o entidades con los siguientes fines:

- Investigadores (personas a cargo del estudio), personal de la investigación, estudiantes a fin de realizar la investigación descrita en el consentimiento informado y otras actividades relacionadas con la investigación, como llevar a cabo análisis de seguridad.
- Los patrocinadores de la investigación, J-PAL North America and the National Bureau of Economic Research, y sus representantes autorizados, socios comerciales, organizaciones de investigación clínica y afiliadas con los fines descritos en el consentimiento informado y para otras actividades relacionadas con la investigación, como la evaluación de la seguridad o la eficacia del medicamento, el dispositivo o tratamiento incluidos en el estudio, la mejora de los diseños de estudios futuros o la obtención de aprobación para nuevos medicamentos, dispositivos o productos de atención de salud.
- Las Juntas de Revisión Institucionales de USC que revisan las investigaciones con seres humanos de conformidad con las regulaciones.
- La organización de ensayos clínicos de USC que respalda la administración de ensayos clínicos en USC.
- Otras oficinas de USC involucradas en cuestiones de cumplimiento de las regulaciones, incluidas las Oficinas del Consejero Jurídico y Cumplimiento.

2

Título del estudio: COVID-19 y Comportamiento de Salud Preventivos

N.° IRB. UP-21-00030

 Entidades gubernamentales de los EE. UU., como la Administración de Medicamentos y Alimentos (FDA, por sus siglas en inglés) y la Oficina para la Protección de los Seres Humanos en la Investigación (OHRP, por sus siglas en inglés), entidades gubernamentales de otros países, y otros que están autorizados por ley a revisar o supervisar esta investigación.

# 5. Creación de una base de datos de investigación:

La actividad de investigación que se presenta a continuación es opcional. Puede elegir si quiere participar o no en estas actividades y su decisión no afectará su capacidad de participar en el estudio de investigación principal. Escriba sus iniciales en la línea que aparece a continuación si desea conceder su permiso específico para esta actividad.

Con frecuencia, los investigadores estudiarán la información de salud existente de grandes grupos de pacientes con el propósito de probar o validar las teorías que desarrolla el investigador. Al escribir sus iniciales más arriba, usted autoriza al equipo de investigación de USC a incluir su información de salud en una base de datos o almacén de investigación con la intención de realizar investigaciones futuras. La Junta de Revisión Institucional de USC puede revisar el modo en que el investigador utiliza o divulga su información de salud para investigaciones futuras.

Esta sección de la autorización permanecerá en vigencia indefinidamente a menos que usted revoque (cancele) esta autorización según se describe a continuación.

# 6. Alcance de esta autorización:

El equipo de investigación de USC solamente puede utilizar y divulgar su información de salud con los fines descritos en esta autorización y en el consentimiento informado o conforme a lo permitido por la ley. Sin embargo, es posible que la información de salud que se comparta con otros ajenos a USC no esté protegida por la ley HIPAA una vez que se haya divulgado. Cierta información de salud puede seguir estando protegida en virtud de la ley estatal.

# 7. Derecho a denegar el acceso a la información de salud:

Es posible que no se le permita consultar (revisar o copiar) su información de salud creada durante este estudio de investigación mientras el estudio de investigación se

Título del estudio: COVID-19 y Comportamiento de Salud Preventivos

N.° IRB. UP-21-00030

esté llevando a cabo. Es posible que tenga derecho a tener acceso a su información de salud una vez que el estudio de investigación haya finalizado.

# 8. Plazo de esta autorización:

Excepto por la búsqueda en la base de datos, esta autorización vence en 25 años a partir de la fecha en que se complete o finalice el estudio.

# 9. Negación a firmar/derecho a revocar:

Debe firmar esta autorización para participar en esta investigación. Usted puede cambiar de parecer y revocar (retirar o cancelar) esta autorización y su participación en este estudio de investigación en cualquier momento. Para hacerlo, su revocación debe enviarse por escrito al Investigador Principal y debe incluir: (1) el título del estudio de investigación; y (2) su nombre y número de teléfono o dirección. Envie la revocación a:

4

Título del estudio: COVID-19 y Comportamiento de Salud Preventivos

N.° IRB. UP-21-00030

Profesora Mireille Jacobson

3715 McClintock Ave

Los Angeles, CA 90089

No se le permitirá participar en la investigación y dejaremos de recopilar su información de salud que le identifique a partir de la fecha en que el Investigador Principal reciba su revocación. Sin embargo, podremos seguir usando y compartiendo la información de salud sobre usted que ya habíamos obtenido según sea necesario para mantener la integridad del estudio de investigación. Además, si la ley lo exige, los investigadores, el patrocinador y las entidades gubernamentales pueden continuar utilizando sus registros para revisar la calidad o la seguridad del estudio.

# 10. Preguntas con respecto a sus derechos de privacidad:

Si tiene preguntas acerca de sus derechos de privacidad, comuníquese con la Oficina de Cumplimiento (Office of Compliance) de USC por teléfono al 213-740-8258 o por correo electrónico a compliance@usc.edu.

# **Consentimiento:**

He leído (u otra persona me leyó) la información que figura más arriba. Me han brindado la oportunidad de hacer preguntas y todas mis preguntas han sido respondidas a mi entera satisfacción. Con mi firma a continuación, acepto que mi información de salud se utilice según se detalla en este formulario.

| Nombre del participante | Firma | Fecha de firma |
|-------------------------|-------|----------------|

5

# **APPENDIX C**: MOP Modifications Log

| Date<br>Modified | Version # | Section #s | Page #s | Brief Summary |
|---|---|---|---|---|
| 06/03/2021 | 1.1 | Section 5.0;<br>Appendix A;<br>Appendix B | Pages 4;<br>48-53; 59-<br>63 | Increase in baseline survey incentive (from \$5 to \$25), to include IRB-approved protocol amendment and revised informed consent documents. |